CLINICAL TRIAL: NCT01128426
Title: Postlicensure Observational Safety Study of 13-valent Pneumococcal Conjugate Vaccine (13vPnC) Administered in Routine Use to Infants and Toddlers
Brief Title: Postlicensure Observational Safety Study of 13vPnC Administered to Infants and Toddlers
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: 6096A1-4002; B1851044
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-06

CONDITIONS: Pneumococcal Disease
Keywords: Pneumococcal conjugate vaccine
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The purpose of the study is to expand the understanding of the safety profile of 13vPnC in routine use following licensure and introduction of the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Infants starting vaccination with 13vPnC in the first 6 months of life who are members of the Northern California Kaiser Permanente healthcase system and who receive at least 1 dose of 13vPnC during the study observation period will be included. Infants must not have had 7vPnC at the time of 13vPnC dose administration.

Exclusion Criteria:

* Infants and children who were previously vaccinated with any number of doses of 7vPnC will be excluded.

Ages: 2 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 60,000 infants total: at least 43,000 infants who receive all 3 primary series doses of 13vPnC plus 15,000 additional infants who receive less than 3 doses of 13vPnC
Sampling Method: Non-Probability Sample
Enrollment: 53902 (Actual)
Dates: Start 2010-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Northern California Kaiser Permanente, Oakland, California, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6096A1-4002&StudyName=Postlicensure%20Observational%20Safety%20Study%20of%2013vPnC%20Administered%20to%20Infants%20and%20Toddlers

RESULTS

PARTICIPANT FLOW:
Groups:
- 13vPnC: Participants enrolled in Kaiser Permanente Northern California (KPNC) health maintenance organization who received 3 primary doses of 13-valent pneumococcal conjugate vaccine (13vPnC, Prevnar 13 or Prevenar 13) within the first 6 months of life at approximately 2, 4, and 6 months of age, according to the Advisory Committee on Immunization Practices (ACIP)-recommended schedule. Participants may also have received fourth dose of 13vPnC according to the ACIP-recommended schedule. Participants were observed for 6 months follow up after Dose 3.
Period: Overall Study
Arm/Group | 13vPnC
Started | 53902
Completed | 53902
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included participants who started vaccination with 13vPnC within the first 6 months of life, were members of KPNC and received at least 1 dose of 13vPnC vaccine during the study observation period.
Arm/Group | 13vPnC
Number analyzed (Participants) | 53902
Age, Continuous [Median (Full Range); unit: days] | 63 [34 to 179]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26274
  Male | 27628

OUTCOME MEASURES:

1. Primary Outcome: Relative Risk of Medically Attended Events Between 30-day Risk Window and 30-day Self-control Window: Pre-Dose 1 Inpatient
Description: Relative risk for given event=incidence rate(risk window)/incidence rate(self-control window).Relative risk in inpatient health care setting for pre-dose 1 assessed by comparing incidence rate of reported events in inpatient setting/1000 person-months occurring within 30 days after Dose 1(30-day risk window) with self-control period occurring during 30 days before Dose 1(pre-vaccination 30-day self-control window).Relative risk,exact 2-sided 90 percent (%) confidence intervals (CIs) reported. Medically attended events documented retrospectively according to International Classification of Diseases, ninth Revision (ICD-9) coding.Medical attended event acute bronchiolitis due to Respiratory Syncytial Virus (RSV) has been represented as acute bronchiolitis due to RSV and acute pyelonephritis without renal medullary necrosis(RMN) lesion has been represented as acute pyelonephritis without RMN lesion in measure categories below.Results reported for events reported in either of the windows.
Time Frame: 30 days before Dose 1 (-34 to -5 days before Dose 1, pre-vaccination self-control window for Dose 1), 30 days after Dose 1 (risk window for Dose 1)
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: ratio
Groups:
- 13vPnC: Participants enrolled in Kaiser Permanente Northern California (KPNC) health maintenance organization who received first primary dose of 13-valent pneumococcal conjugate vaccine (13vPnC, Prevnar 13 or Prevenar 13) within the first 6 months of life at approximately 2 months of age, according to the Advisory Committee on Immunization Practices (ACIP)-recommended schedule.
Arm/Group | 13vPnC
Number analyzed (Participants) | 53902
ratio
  Abnormal involuntary movements | 0.98 [0.23 to 4.21]
  Acute bronchiolitis due to RSV | 0.46 [0.32 to 0.66]
  Acute febrile mucocutaneous lymph node syndrome | 0.98 [0.05 to 18.69]
  Acute otitis media | 0.30 [0.09 to 0.85]
  Acute pyelonephritis without RMN lesion | 0.49 [0.19 to 1.21]
  Alkalosis | 1.18 [0.42 to 3.38]
  Apnea | 0.55 [0.27 to 1.10]
  Apparent life threatening event infant | 0.45 [0.24 to 0.82]
  Asthma, unspecified, unspecified status | NA [1.68 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Bronchiolitis | 0.51 [0.29 to 0.89]
  Bronchitis | NA [0.11 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Bronchospasm | NA [NA to 8.85] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Candidiasis of mouth | 0.53 [0.24 to 1.14]
  Cellulitis and abscess of trunk | 0.98 [0.23 to 4.21]
  Constipation | 0.25 [0.02 to 1.46]
  Croup | NA [1.68 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Dehydration | 0.49 [0.30 to 0.80]
  Dermatitis | 0.25 [0.02 to 1.46]
  Dyspnea | 0.68 [0.32 to 1.40]
  Failure to thrive | 0.87 [0.49 to 1.55]
  Fever | 0.28 [0.17 to 0.45]
  Fussy infant | 0.49 [0.13 to 1.59]
  Gastroenteritis | NA [NA to 0.58] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Hypopotassemia | 0.66 [0.12 to 3.21]
  Lipoma of other specified sites | NA [0.11 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Methicillin susceptible Staphylococcus aureus | 1.64 [0.48 to 6.20]
  Nausea and vomiting | NA [NA to 8.85] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Neonatal bradycardia | 0.18 [0.07 to 0.42]
  Neonatal candida infection | NA [NA to 0.58] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Other diseases of nasal cavity and sinuses | 0.49 [0.16 to 1.35]
  Other specified cardiac dysrhythmias | 0.98 [0.40 to 2.44]
  Pilonidal cyst without mention of abscess | 7.22 [3.64 to 15.68]
  Pneumonia | 0.41 [0.16 to 0.97]
  Primary apnea of newborn | 0.13 [0.06 to 0.28]
  Rash | 0.22 [0.05 to 0.75]
  Respiratory syncytial virus | 0.12 [0.01 to 0.61]
  Retinopathy of prematurity stage 2 | 0.74 [0.19 to 2.75]
  Single seizure | 1.12 [0.47 to 2.72]
  Stridor | 0.79 [0.24 to 2.48]
  Umbilical hernia without obstruction/gangrene | 0.49 [0.26 to 0.90]
  Unspecified bacterial pneumonia | 3.93 [0.66 to 48.16]
  Unspecified septicemia | 1.18 [0.42 to 3.38]
  Urinary tract infection | 0.23 [0.12 to 0.43]
  Viral syndrome | 0.41 [0.19 to 0.84]
  Weakness | NA [0.45 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
Statistical Analysis 1: Comparison: 13vPnC; Abnormal involuntary movements: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.98, mid-p exact binomial method
Statistical Analysis 2: Comparison: 13vPnC; Acute bronchiolitis due to RSV: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 3: Comparison: 13vPnC; Acute febrile mucocutaneous lymph node syndrome: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0 .99, mid-p exact binomial method
Statistical Analysis 4: Comparison: 13vPnC; Acute otitis media: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.05, mid-p exact binomial method
Statistical Analysis 5: Comparison: 13vPnC; Acute pyelonephritis without RMN lesion: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0 .20, mid-p exact binomial method
Statistical Analysis 6: Comparison: 13vPnC; Alkalosis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.79, mid-p exact binomial method
Statistical Analysis 7: Comparison: 13vPnC; Apnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.16, mid-p exact binomial method
Statistical Analysis 8: Comparison: 13vPnC; Apparent life threatening event infant: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.03, mid-p exact binomial method
Statistical Analysis 9: Comparison: 13vPnC; Asthma, unspecified, unspecified status: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0 .03, mid-p exact binomial method
Statistical Analysis 10: Comparison: 13vPnC; Bronchiolitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.05, mid-p exact binomial method
Statistical Analysis 11: Comparison: 13vPnC; Bronchitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 12: Comparison: 13vPnC; Bronchospasm: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 13: Comparison: 13vPnC; Candidiasis of mouth: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.18, mid-p exact binomial method
Statistical Analysis 14: Comparison: 13vPnC; Cellulitis and abscess of trunk: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.98, mid-p exact binomial method
Statistical Analysis 15: Comparison: 13vPnC; Constipation: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.21, mid-p exact binomial method
Statistical Analysis 16: Comparison: 13vPnC; Croup: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.03, mid-p exact binomial method
Statistical Analysis 17: Comparison: 13vPnC; Dehydration: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.01, mid-p exact binomial method
Statistical Analysis 18: Comparison: 13vPnC; Dermatitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.21, mid-p exact binomial method
Statistical Analysis 19: Comparison: 13vPnC; Dyspnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.38, mid-p exact binomial method
Statistical Analysis 20: Comparison: 13vPnC; Failure to thrive: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.70, mid-p exact binomial method
Statistical Analysis 21: Comparison: 13vPnC; Fever: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 22: Comparison: 13vPnC; Fussy infant: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.33, mid-p exact binomial method
Statistical Analysis 23: Comparison: 13vPnC; Gastroenteritis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.03, mid-p exact binomial method
Statistical Analysis 24: Comparison: 13vPnC; Hypopotassemia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.67, mid-p exact binomial method
Statistical Analysis 25: Comparison: 13vPnC; Lipoma of other specified sites: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 26: Comparison: 13vPnC; Methicillin susceptible Staphylococcus aureus: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 27: Comparison: 13vPnC; Nausea and vomiting: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 28: Comparison: 13vPnC; Neonatal bradycardia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 29: Comparison: 13vPnC; Neonatal candida infection: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.03, mid-p exact binomial method
Statistical Analysis 30: Comparison: 13vPnC; Other diseases of nasal cavity and sinuses: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.26, mid-p exact binomial method
Statistical Analysis 31: Comparison: 13vPnC; Other specified cardiac dysrhythmias: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.98, mid-p exact binomial method
Statistical Analysis 32: Comparison: 13vPnC; Pilonidal cyst without mention of abscess: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 33: Comparison: 13vPnC; Pneumonia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.09, mid-p exact binomial method
Statistical Analysis 34: Comparison: 13vPnC; Primary apnea of newborn: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 35: Comparison: 13vPnC; Rash: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.04, mid-p exact binomial method
Statistical Analysis 36: Comparison: 13vPnC; Respiratory syncytial virus: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.02, mid-p exact binomial method
Statistical Analysis 37: Comparison: 13vPnC; Retinopathy of prematurity stage 2: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.71, mid-p exact binomial method
Statistical Analysis 38: Comparison: 13vPnC; Single seizure: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.83, mid-p exact binomial method
Statistical Analysis 39: Comparison: 13vPnC; Stridor: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.74, mid-p exact binomial method
Statistical Analysis 40: Comparison: 13vPnC; Umbilical hernia without obstruction/gangrene: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.05, mid-p exact binomial method
Statistical Analysis 41: Comparison: 13vPnC; Unspecified bacterial pneumonia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.23, mid-p exact binomial method
Statistical Analysis 42: Comparison: 13vPnC; Unspecified septicemia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.79, mid-p exact binomial method
Statistical Analysis 43: Comparison: 13vPnC; Urinary tract infection: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 44: Comparison: 13vPnC; Viral syndrome: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.04, mid-p exact binomial method
Statistical Analysis 45: Comparison: 13vPnC; Weakness: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.25, mid-p exact binomial method

2. Primary Outcome: Relative Risk of Medically Attended Events Between 30-day Risk Window and 30-day Self-control Window: Pre-Dose 1 Emergency Department
Description: Relative risk for given event = incidence rate (risk window) / incidence rate (self-control window). Relative risk in emergency department health care setting for pre-dose 1 was assessed by comparing the incidence rate of reported events in emergency department setting per 1000 person-months occurring within 30 days after Dose 1 (30-day risk window) with self-control period occurring during 30 days before Dose 1 (pre-vaccination 30-day self-control window). Relative risk and exact 2-sided 90% CIs were reported. Medically attended events were documented retrospectively according to ICD-9 coding. Results were reported for events reported in either of the windows.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: ratio
Arm/Group | 13vPnC
Number analyzed (Participants) | 53902
ratio
  Abnormal involuntary movements | 1.97 [0.23 to 28.51]
  Acute bronchiolitis due to RSV | 0.27 [0.12 to 0.56]
  Acute otitis media | 2.75 [1.19 to 6.96]
  Acute pyelonephritis without RMN lesion | NA [NA to 8.85] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Adverse drug reaction | 0.98 [0.05 to 18.69]
  Alkalosis | NA [0.11 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Apnea | 0.77 [0.32 to 1.78]
  Apparent life threatening event infant | 0.72 [0.37 to 1.39]
  Asthma with acute exacerbation | NA [0.11 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Asthma, unspecified, unspecified status | 0.74 [0.19 to 2.75]
  Bronchiolitis | 0.82 [0.57 to 1.17]
  Bronchitis | 0.33 [0.03 to 2.20]
  Bronchospasm | 2.95 [0.79 to 14.40]
  Candidiasis of mouth | 0.14 [0.03 to 0.45]
  Constipation | 0.36 [0.17 to 0.70]
  Croup | 12.79 [2.78 to 136.60]
  Dehydration | 0.84 [0.32 to 2.16]
  Dermatitis | 0.36 [0.12 to 0.92]
  Dyspnea | 0.77 [0.45 to 1.29]
  Failure to thrive | 1.97 [0.23 to 28.51]
  Fever | 0.57 [0.48 to 0.68]
  Fussy infant | 0.67 [0.48 to 0.92]
  Gastroenteritis | 0.82 [0.29 to 2.29]
  Hematoma | 0.98 [0.05 to 18.69]
  Methicillin susceptible Staphylococcus aureus | NA [NA to 8.85] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Nausea and vomiting | 0.45 [0.31 to 0.65]
  Neonatal candida infection | 0.18 [0.04 to 0.59]
  Other diseases of nasal cavity and sinuses | 0.27 [0.18 to 0.42]
  Other specified cardiac dysrhythmias | NA [NA to 1.14] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Pneumonia | 0.93 [0.52 to 1.65]
  Primary apnea of newborn | NA [NA to 1.14] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Rash | 0.70 [0.41 to 1.17]
  Respiratory syncytial virus | 1.12 [0.47 to 2.72]
  Single seizure | 0.98 [0.37 to 2.64]
  Stomatitis | NA [NA to 8.85] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Stridor | NA [NA to 0.77] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Subconjunctival hemorrhage | 1.97 [0.23 to 28.51]
  Umbilical hernia without obstruction/gangrene | 0.14 [0.03 to 0.45]
  Unspecified septicemia | 0.79 [0.24 to 2.48]
  Urinary tract infection | 0.89 [0.58 to 1.36]
  Urticaria | NA [0.85 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Vaccines adverse reaction | NA [0.85 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Viral syndrome | 0.83 [0.51 to 1.34]
  Weakness | 0.49 [0.03 to 4.23]
  Wheezing | 0.84 [0.32 to 2.16]
Statistical Analysis 1: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.63, mid-p exact binomial method
Statistical Analysis 2: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 3: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p = 0.04, mid-p exact binomial method
Statistical Analysis 4: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 5: Comparison: 13vPnC; Adverse drug reaction: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.99, mid-p exact binomial method
Statistical Analysis 6: Comparison: 13vPnC; Alkalosis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 7: Comparison: 13vPnC; Apnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.61, mid-p exact binomial method
Statistical Analysis 8: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; p = 0.42, mid-p exact binomial method
Statistical Analysis 9: Comparison: 13vPnC; Asthma with acute exacerbation: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 10: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; p = 0.71, mid-p exact binomial method
Statistical Analysis 11: Comparison: 13vPnC; Bronchiolitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.36, mid-p exact binomial method
Statistical Analysis 12: Comparison: 13vPnC; Bronchitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.37, mid-p exact binomial method
Statistical Analysis 13: Comparison: 13vPnC; Bronchospasm: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.19, mid-p exact binomial method
Statistical Analysis 14: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 15: Comparison: 13vPnC; Constipation: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 16: Comparison: 13vPnC; Croup: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 17: Comparison: 13vPnC; Dehydration: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.77, mid-p exact binomial method
Statistical Analysis 18: Comparison: 13vPnC; Dermatitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.07, mid-p exact binomial method
Statistical Analysis 19: Comparison: 13vPnC; Dyspnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.41, mid-p exact binomial method
Statistical Analysis 20: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 20]; Test type: Superiority or Other; p = 0.63, mid-p exact binomial method
Statistical Analysis 21: Comparison: 13vPnC; Fever: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 22: Comparison: 13vPnC; Fussy infant: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.04, mid-p exact binomial method
Statistical Analysis 23: Comparison: 13vPnC; Gastroenteritis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.75, mid-p exact binomial method
Statistical Analysis 24: Comparison: 13vPnC; Hematoma: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.99, mid-p exact binomial method
Statistical Analysis 25: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 26]; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 26: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 27]; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 27: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 29]; Test type: Superiority or Other; p = 0.01, mid-p exact binomial method
Statistical Analysis 28: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 30]; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 29: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 31]; Test type: Superiority or Other; p = 0.12, mid-p exact binomial method
Statistical Analysis 30: Comparison: 13vPnC; Pneumonia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.83, mid-p exact binomial method
Statistical Analysis 31: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 34]; Test type: Superiority or Other; p = 0.12, mid-p exact binomial method
Statistical Analysis 32: Comparison: 13vPnC; Rash: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.26, mid-p exact binomial method
Statistical Analysis 33: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 36]; Test type: Superiority or Other; p = 0.83, mid-p exact binomial method
Statistical Analysis 34: Comparison: 13vPnC; Single seizure: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.98, mid-p exact binomial method
Statistical Analysis 35: Comparison: 13vPnC; Stomatitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 36: Comparison: 13vPnC; Stridor: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.06, mid-p exact binomial method
Statistical Analysis 37: Comparison: 13vPnC; Subconjunctival hemorrhage: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.63, mid-p exact binomial method
Statistical Analysis 38: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 40]; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 39: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 42]; Test type: Superiority or Other; p = 0.74, mid-p exact binomial method
Statistical Analysis 40: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 43]; Test type: Superiority or Other; p = 0.66, mid-p exact binomial method
Statistical Analysis 41: Comparison: 13vPnC; Urticaria: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.13, mid-p exact binomial method
Statistical Analysis 42: Comparison: 13vPnC; Vaccines adverse reaction: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.13, mid-p exact binomial method
Statistical Analysis 43: Comparison: 13vPnC; Viral syndrome: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.53, mid-p exact binomial method
Statistical Analysis 44: Comparison: 13vPnC; Weakness: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.62, mid-p exact binomial method
Statistical Analysis 45: Comparison: 13vPnC; Wheezing: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.77, mid-p exact binomial method

3. Primary Outcome: Relative Risk of Medically Attended Events Between 30-day Risk Window and 30-day Self-control Window: Pre-Dose 1 Inpatient and Emergency Department Combined
Description: Relative risk for given event = incidence rate (risk window) / incidence rate (self-control window). Relative risk in inpatient and emergency department health care setting for pre-dose 1 was assessed by comparing the overall incidence rates of reported events in both settings per 1000 person-months occurring within 30 days after Dose 1 (30-day risk window) with self-control period occurring during 30 days before Dose 1 (pre-vaccination 30-day self-control window). Relative risk and exact 2-sided 90% CIs were reported. Medically attended events were documented retrospectively according to ICD-9 coding. Results were reported for events reported in either of the windows.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: ratio
Arm/Group | 13vPnC
Number analyzed (Participants) | 53902
ratio
  Abnormal involuntary movements | 1.23 [0.39 to 4.01]
  Acute bronchiolitis due to RSV | 0.45 [0.32 to 0.63]
  Acute febrile mucocutaneous lymph node syndrome | 0.98 [0.05 to 18.69]
  Acute otitis media | 1.19 [0.66 to 2.19]
  Acute pyelonephritis without RMN lesion | 0.49 [0.19 to 1.21]
  Adverse drug reaction | 0.98 [0.05 to 18.69]
  Alkalosis | 1.18 [0.42 to 3.38]
  Apnea | 0.56 [0.31 to 0.98]
  Apparent life threatening event infant | 0.51 [0.30 to 0.84]
  Asthma with acute exacerbation | NA [0.11 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Asthma, unspecified, unspecified status | 1.72 [0.61 to 5.26]
  Bronchiolitis | 0.71 [0.52 to 0.96]
  Bronchitis | 0.66 [0.12 to 3.21]
  Bronchospasm | 1.97 [0.61 to 7.19]
  Candidiasis of mouth | 0.37 [0.19 to 0.69]
  Cellulitis and abscess of trunk | 0.98 [0.23 to 4.21]
  Constipation | 0.34 [0.17 to 0.64]
  Croup | 13.77 [3.02 to 146.40]
  Dehydration | 0.55 [0.35 to 0.86]
  Dermatitis | 0.35 [0.14 to 0.82]
  Dyspnea | 0.78 [0.50 to 1.19]
  Failure to thrive | 0.88 [0.50 to 1.53]
  Fever | 0.57 [0.48 to 0.67]
  Fussy infant | 0.64 [0.46 to 0.87]
  Gastroenteritis | 0.45 [0.17 to 1.08]
  Hematoma | 0.98 [0.05 to 18.69]
  Hypopotassemia | 0.66 [0.12 to 3.21]
  Lipoma of other specified sites | NA [0.11 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Methicillin susceptible Staphylococcus aureus | 1.23 [0.39 to 4.01]
  Nausea and vomiting | 0.45 [0.31 to 0.65]
  Neonatal bradycardia | 0.18 [0.07 to 0.42]
  Neonatal candida infection | 0.12 [0.03 to 0.39]
  Other diseases of nasal cavity and sinuses | 0.30 [0.20 to 0.44]
  Other specified cardiac dysrhythmias | 0.77 [0.32 to 1.78]
  Pilonidal cyst without mention of abscess | 7.22 [3.64 to 15.68]
  Pneumonia | 0.74 [0.44 to 1.23]
  Primary apnea of newborn | 0.12 [0.05 to 0.26]
  Rash | 0.57 [0.35 to 0.91]
  Respiratory syncytial virus | 0.68 [0.32 to 1.40]
  Retinopathy of prematurity stage 2 | 0.74 [0.19 to 2.75]
  Single seizure | 0.98 [0.51 to 1.90]
  Stomatitis | NA [NA to 8.85] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Stridor | 0.49 [0.16 to 1.35]
  Subconjunctival hemorrhage | 1.97 [0.23 to 28.51]
  Umbilical hernia without obstruction/gangrene | 0.38 [0.22 to 0.64]
  Unspecified bacterial pneumonia | 3.93 [0.66 to 48.16]
  Unspecified septicemia | 1.09 [0.51 to 2.38]
  Urinary tract infection | 0.59 [0.41 to 0.85]
  Urticaria | NA [0.85 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Vaccines adverse reaction | NA [0.85 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Viral syndrome | 0.66 [0.44 to 0.98]
  Weakness | 0.98 [0.15 to 6.28]
  Wheezing | 0.84 [0.32 to 2.16]
Statistical Analysis 1: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.77, mid-p exact binomial method
Statistical Analysis 2: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 3: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.99, mid-p exact binomial method
Statistical Analysis 4: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p = 0.63, mid-p exact binomial method
Statistical Analysis 5: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.20, mid-p exact binomial method
Statistical Analysis 6: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.99, mid-p exact binomial method
Statistical Analysis 7: Comparison: 13vPnC; Alkalosis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.79, mid-p exact binomial method
Statistical Analysis 8: Comparison: 13vPnC; Apnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.09, mid-p exact binomial method
Statistical Analysis 9: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; p = 0.03, mid-p exact binomial method
Statistical Analysis 10: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 11: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; p = 0.40, mid-p exact binomial method
Statistical Analysis 12: Comparison: 13vPnC; Bronchiolitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.07, mid-p exact binomial method
Statistical Analysis 13: Comparison: 13vPnC; Bronchitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.67, mid-p exact binomial method
Statistical Analysis 14: Comparison: 13vPnC; Bronchospasm: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.36, mid-p exact binomial method
Statistical Analysis 15: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 16: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 14]; Test type: Superiority or Other; p = 0.98, mid-p exact binomial method
Statistical Analysis 17: Comparison: 13vPnC; Constipation: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 18: Comparison: 13vPnC; Croup: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 19: Comparison: 13vPnC; Dehydration: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.03, mid-p exact binomial method
Statistical Analysis 20: Comparison: 13vPnC; Dermatitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.04, mid-p exact binomial method
Statistical Analysis 21: Comparison: 13vPnC; Dyspnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.33, mid-p exact binomial method
Statistical Analysis 22: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 20]; Test type: Superiority or Other; p = 0.71, mid-p exact binomial method
Statistical Analysis 23: Comparison: 13vPnC; Fever: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 24: Comparison: 13vPnC; Fussy infant: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.02, mid-p exact binomial method
Statistical Analysis 25: Comparison: 13vPnC; Gastroenteritis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.13, mid-p exact binomial method
Statistical Analysis 26: Comparison: 13vPnC; Hematoma: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.99, mid-p exact binomial method
Statistical Analysis 27: Comparison: 13vPnC; Hypopotassemia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.67, mid-p exact binomial method
Statistical Analysis 28: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 25]; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 29: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 26]; Test type: Superiority or Other; p = 0.77, mid-p exact binomial method
Statistical Analysis 30: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 27]; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 31: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 28]; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 32: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 29]; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 33: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 30]; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 34: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 31]; Test type: Superiority or Other; p = 0.61, mid-p exact binomial method
Statistical Analysis 35: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 32]; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 36: Comparison: 13vPnC; Pneumonia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.33, mid-p exact binomial method
Statistical Analysis 37: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 34]; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 38: Comparison: 13vPnC; Rash: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.05, mid-p exact binomial method
Statistical Analysis 39: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 36]; Test type: Superiority or Other; p = 0.38, mid-p exact binomial method
Statistical Analysis 40: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 37]; Test type: Superiority or Other; p = 0.71, mid-p exact binomial method
Statistical Analysis 41: Comparison: 13vPnC; Single seizure: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.97, mid-p exact binomial method
Statistical Analysis 42: Comparison: 13vPnC; Stomatitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 43: Comparison: 13vPnC; Stridor: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.26, mid-p exact binomial method
Statistical Analysis 44: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 37]; Test type: Superiority or Other; p = 0.63, mid-p exact binomial method
Statistical Analysis 45: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 40]; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 46: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 41]; Test type: Superiority or Other; p = 0.23, mid-p exact binomial method
Statistical Analysis 47: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 42]; Test type: Superiority or Other; p = 0.85, mid-p exact binomial method
Statistical Analysis 48: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 43]; Test type: Superiority or Other; p = 0.02, mid-p exact binomial method
Statistical Analysis 49: Comparison: 13vPnC; Urticaria: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.13, mid-p exact binomial method
Statistical Analysis 50: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 42]; Test type: Superiority or Other; p = 0.13, mid-p exact binomial method
Statistical Analysis 51: Comparison: 13vPnC; Viral syndrome: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.09, mid-p exact binomial method
Statistical Analysis 52: Comparison: 13vPnC; Weakness: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.99, mid-p exact binomial method
Statistical Analysis 53: Comparison: 13vPnC; Wheezing: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.77, mid-p exact binomial method

4. Primary Outcome: Relative Risk of Medically Attended Events Between 30-day Risk Window and 30-day Self-control Window: Dose 1 Inpatient
Description: Relative risk for given event = incidence rate (risk window) / incidence rate (self-control window). Relative risk in inpatient health care setting for Dose 1 was assessed by comparing the incidence rate of reported events in inpatient setting per 1000 person-months occurring within 30 days after Dose 1 (30-day risk window) with the self-control period occurring during the subsequent 30 days (30-day self-control window). Relative risk and exact 2-sided 90% (CIs were reported. Medically attended events were documented retrospectively according to ICD-9 coding. Results were reported for events reported in either of the windows.
Time Frame: 30 days after Dose 1 (risk window for Dose 1), 30 days after risk window (post-dose self-control window for Dose 1)
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: ratio
Arm/Group | 13vPnC
Number analyzed (Participants) | 53902
ratio
  Abnormal involuntary movements | NA [0.79 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Acute bronchiolitis due to RSV | 2.65 [1.51 to 4.83]
  Acute febrile mucocutaneous lymph node syndrome | 0.91 [0.05 to 17.29]
  Acute otitis media | 0.91 [0.21 to 3.90]
  Acute pyelonephritis without RMN lesion | 1.14 [0.36 to 3.71]
  Alkalosis | NA [1.95 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Apnea | 2.73 [0.93 to 9.39]
  Apparent life threatening event infant | 2.50 [0.97 to 7.18]
  Asthma, unspecified, unspecified status | NA [1.56 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Bronchiolitis | 1.69 [0.78 to 3.81]
  Bronchitis | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Candidiasis of mouth | 6.37 [1.26 to 71.83]
  Cellulitis and abscess of trunk | 2.73 [0.41 to 35.48]
  Constipation | 0.30 [0.02 to 2.03]
  Croup | 0.91 [0.31 to 2.71]
  Dehydration | 1.11 [0.61 to 2.03]
  Dermatitis | 0.46 [0.03 to 3.92]
  Dyspnea | 2.05 [0.77 to 6.03]
  Failure to thrive | 1.62 [0.82 to 3.31]
  Fever | 1.95 [0.92 to 4.32]
  Fussy infant | 2.73 [0.41 to 35.48]
  Gastroenteritis | NA [NA to 1.97] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Hypopotassemia | NA [0.42 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Lipoma of other specified sites | 0.46 [0.03 to 3.92]
  Methicillin susceptible Staphylococcus aureus | 4.55 [0.83 to 53.66]
  Nausea and vomiting | NA [NA to 8.19] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Neonatal bradycardia | NA [1.17 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Other diseases of nasal cavity and sinuses | 0.61 [0.19 to 1.80]
  Other specified cardiac dysrhythmias | 3.19 [0.88 to 15.19]
  Pilonidal cyst without mention of abscess | 2.36 [1.48 to 3.83]
  Pneumonia | 0.91 [0.31 to 2.17]
  Primary apnea of newborn | NA [1.56 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Rash | 0.91 [0.14 to 5.82]
  Respiratory syncytial virus | 0.91 [0.05 to 17.29]
  Retinopathy of prematurity stage 2 | NA [0.79 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Single seizure | 0.66 [0.30 to 1.43]
  Stridor | 0.91 [0.26 to 3.13]
  Umbilical hernia without obstruction/gangrene | 2.50 [0.97 to 7.18]
  Unspecified bacterial pneumonia | NA [1.17 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Unspecified septicemia | 5.46 [1.04 to 62.75]
  Urinary tract infection | 1.82 [0.66 to 5.45]
  Viral syndrome | 1.06 [0.41 to 2.77]
  Weakness | NA [0.42 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
Statistical Analysis 1: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.14, mid-p exact binomial method
Statistical Analysis 2: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 3: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.95, mid-p exact binomial method
Statistical Analysis 4: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p = 0.91, mid-p exact binomial method
Statistical Analysis 5: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.86, mid-p exact binomial method
Statistical Analysis 6: Comparison: 13vPnC; Alkalosis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.02, mid-p exact binomial method
Statistical Analysis 7: Comparison: 13vPnC; Apnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.13, mid-p exact binomial method
Statistical Analysis 8: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; p = 0.11, mid-p exact binomial method
Statistical Analysis 9: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; p = 0.04, mid-p exact binomial method
Statistical Analysis 10: Comparison: 13vPnC; Bronchiolitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.27, mid-p exact binomial method
Statistical Analysis 11: Comparison: 13vPnC; Bronchitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 12: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; p = 0.05, mid-p exact binomial method
Statistical Analysis 13: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 14]; Test type: Superiority or Other; p = 0.42, mid-p exact binomial method
Statistical Analysis 14: Comparison: 13vPnC; Constipation: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.33, mid-p exact binomial method
Statistical Analysis 15: Comparison: 13vPnC; Croup: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.88, mid-p exact binomial method
Statistical Analysis 16: Comparison: 13vPnC; Dehydration: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.79, mid-p exact binomial method
Statistical Analysis 17: Comparison: 13vPnC; Dermatitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.57, mid-p exact binomial method
Statistical Analysis 18: Comparison: 13vPnC; Dyspnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.24, mid-p exact binomial method
Statistical Analysis 19: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 20]; Test type: Superiority or Other; p = 0.25, mid-p exact binomial method
Statistical Analysis 20: Comparison: 13vPnC; Fever: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.14, mid-p exact binomial method
Statistical Analysis 21: Comparison: 13vPnC; Fussy infant: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.42, mid-p exact binomial method
Statistical Analysis 22: Comparison: 13vPnC; Gastroenteritis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.23, mid-p exact binomial method
Statistical Analysis 23: Comparison: 13vPnC; Hypopotassemia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.27, mid-p exact binomial method
Statistical Analysis 24: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 25]; Test type: Superiority or Other; p = 0.57, mid-p exact binomial method
Statistical Analysis 25: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 26]; Test type: Superiority or Other; p = 0.15, mid-p exact binomial method
Statistical Analysis 26: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 27]; Test type: Superiority or Other; p = 0.48, mid-p exact binomial method
Statistical Analysis 27: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 28]; Test type: Superiority or Other; p = 0.08, mid-p exact binomial method
Statistical Analysis 28: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 30]; Test type: Superiority or Other; p = 0.46, mid-p exact binomial method
Statistical Analysis 29: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 31]; Test type: Superiority or Other; p = 0.14, mid-p exact binomial method
Statistical Analysis 30: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 32]; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 31: Comparison: 13vPnC; Pneumonia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.88, mid-p exact binomial method
Statistical Analysis 32: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 34]; Test type: Superiority or Other; p = 0.04, mid-p exact binomial method
Statistical Analysis 33: Comparison: 13vPnC; Rash: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.93, mid-p exact binomial method
Statistical Analysis 34: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 36]; Test type: Superiority or Other; p = 0.95, mid-p exact binomial method
Statistical Analysis 35: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 37]; Test type: Superiority or Other; p = 0.14, mid-p exact binomial method
Statistical Analysis 36: Comparison: 13vPnC; Single seizure: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.38, mid-p exact binomial method
Statistical Analysis 37: Comparison: 13vPnC; Stridor: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.90, mid-p exact binomial method
Statistical Analysis 38: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 40]; Test type: Superiority or Other; p = 0.11, mid-p exact binomial method
Statistical Analysis 39: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 41]; Test type: Superiority or Other; p = 0.08, mid-p exact binomial method
Statistical Analysis 40: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 42]; Test type: Superiority or Other; p = 0.09, mid-p exact binomial method
Statistical Analysis 41: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 43]; Test type: Superiority or Other; p = 0.34, mid-p exact binomial method
Statistical Analysis 42: Comparison: 13vPnC; Viral syndrome: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.92, mid-p exact binomial method
Statistical Analysis 43: Comparison: 13vPnC; Weakness: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.27, mid-p exact binomial method

5. Primary Outcome: Relative Risk of Medically Attended Events Between 30-day Risk Window and 30-day Self-control Window: Dose 1 Emergency Department
Description: Relative risk for given event = incidence rate (risk window) / incidence rate (self-control window). Relative risk in emergency department health care setting for Dose 1 was assessed by comparing the incidence rate of reported events in emergency department setting per 1000 person-months occurring within 30 days after Dose 1 (30-day risk window) with the self-control period occurring during the subsequent 30 days (30-day self-control window). Relative risk and exact 2-sided 90% CIs were reported. Medically attended events were documented retrospectively according to ICD-9 coding. Results were reported for events reported in either of the windows.
Time Frame: 30 days after Dose 1 (risk window for Dose 1), 30 days after risk window (post-dose self-control window for Dose 1)
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: ratio
Arm/Group | 13vPnC
Number analyzed (Participants) | 53902
ratio
  Abnormal involuntary movements | 0.61 [0.11 to 2.97]
  Acute bronchiolitis due to RSV | 0.68 [0.27 to 1.69]
  Acute otitis media | 0.61 [0.34 to 1.07]
  Adverse drug reaction | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Alkalosis | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Apnea | 3.19 [0.88 to 15.19]
  Apparent life threatening event infant | 2.50 [0.97 to 7.18]
  Asthma with acute exacerbation | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Asthma, unspecified, unspecified status | 0.23 [0.07 to 0.63]
  Bronchiolitis | 0.66 [0.47 to 0.93]
  Bronchitis | 0.91 [0.05 to 17.29]
  Bronchospasm | 0.61 [0.24 to 1.46]
  Candidiasis of mouth | 1.82 [0.21 to 26.39]
  Constipation | 0.73 [0.32 to 1.61]
  Croup | 0.59 [0.32 to 1.06]
  Dehydration | 0.61 [0.24 to 1.46]
  Dermatitis | 0.26 [0.09 to 0.64]
  Dyspnea | 1.49 [0.79 to 2.86]
  Failure to thrive | NA [0.42 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Fever | 1.38 [1.11 to 1.72]
  Fussy infant | 1.19 [0.81 to 1.77]
  Gastroenteritis | 0.76 [0.26 to 2.12]
  Hand, foot and mouth disease | NA [NA to 8.19] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Hematoma | 0.91 [0.05 to 17.29]
  Nausea and vomiting | 0.71 [0.47 to 1.07]
  Neonatal candida infection | 1.82 [0.21 to 26.39]
  Other diseases of nasal cavity and sinuses | 0.69 [0.42 to 1.14]
  Other specified cardiac dysrhythmias | NA [NA to 8.19] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Pneumonia | 0.61 [0.35 to 1.03]
  Rash | 0.97 [0.54 to 1.73]
  Respiratory syncytial virus | 3.64 [1.04 to 17.06]
  Single seizure | 0.91 [0.34 to 2.45]
  Stridor | NA [NA to 8.19] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Subconjunctival hemorrhage | NA [0.42 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Umbilical hernia without obstruction/gangrene | 1.82 [0.21 to 26.39]
  Unspecified septicemia | 1.82 [0.42 to 9.58]
  Urinary tract infection | 3.30 [1.74 to 6.62]
  Urticaria | 0.91 [0.21 to 3.90]
  Vaccines adverse reaction | NA [0.79 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Viral syndrome | 0.56 [0.35 to 0.87]
  Weakness | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Wheezing | 0.55 [0.22 to 1.28]
Statistical Analysis 1: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.62, mid-p exact binomial method
Statistical Analysis 2: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.49, mid-p exact binomial method
Statistical Analysis 3: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p = 0.15, mid-p exact binomial method
Statistical Analysis 4: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 5: Comparison: 13vPnC; Alkalosis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 6: Comparison: 13vPnC; Apnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.14, mid-p exact binomial method
Statistical Analysis 7: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; p = 0.11, mid-p exact binomial method
Statistical Analysis 8: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 9: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; p = 0.01, mid-p exact binomial method
Statistical Analysis 10: Comparison: 13vPnC; Bronchiolitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.05, mid-p exact binomial method
Statistical Analysis 11: Comparison: 13vPnC; Bronchitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.95, mid-p exact binomial method
Statistical Analysis 12: Comparison: 13vPnC; Bronchospasm: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.35, mid-p exact binomial method
Statistical Analysis 13: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; p = 0.68, mid-p exact binomial method
Statistical Analysis 14: Comparison: 13vPnC; Constipation: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.51, mid-p exact binomial method
Statistical Analysis 15: Comparison: 13vPnC; Croup: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.14, mid-p exact binomial method
Statistical Analysis 16: Comparison: 13vPnC; Dehydration: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.35, mid-p exact binomial method
Statistical Analysis 17: Comparison: 13vPnC; Dermatitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.01, mid-p exact binomial method
Statistical Analysis 18: Comparison: 13vPnC; Dyspnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.30, mid-p exact binomial method
Statistical Analysis 19: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 20]; Test type: Superiority or Other; p = 0.27, mid-p exact binomial method
Statistical Analysis 20: Comparison: 13vPnC; Fever: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.02, mid-p exact binomial method
Statistical Analysis 21: Comparison: 13vPnC; Fussy infant: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.45, mid-p exact binomial method
Statistical Analysis 22: Comparison: 13vPnC; Gastroenteritis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.66, mid-p exact binomial method
Statistical Analysis 23: Comparison: 13vPnC; Hand, foot and mouth disease: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.48, mid-p exact binomial method
Statistical Analysis 24: Comparison: 13vPnC; Hematoma: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.95, mid-p exact binomial method
Statistical Analysis 25: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 27]; Test type: Superiority or Other; p = 0.17, mid-p exact binomial method
Statistical Analysis 26: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 29]; Test type: Superiority or Other; p = 0.68, mid-p exact binomial method
Statistical Analysis 27: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 30]; Test type: Superiority or Other; p = 0.23, mid-p exact binomial method
Statistical Analysis 28: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 31]; Test type: Superiority or Other; p = 0.48, mid-p exact binomial method
Statistical Analysis 29: Comparison: 13vPnC; Pneumonia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.12, mid-p exact binomial method
Statistical Analysis 30: Comparison: 13vPnC; Rash: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.92, mid-p exact binomial method
Statistical Analysis 31: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 36]; Test type: Superiority or Other; p = 0.09, mid-p exact binomial method
Statistical Analysis 32: Comparison: 13vPnC; Single seizure: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.87, mid-p exact binomial method
Statistical Analysis 33: Comparison: 13vPnC; Stridor: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.48, mid-p exact binomial method
Statistical Analysis 34: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 37]; Test type: Superiority or Other; p = 0.27, mid-p exact binomial method
Statistical Analysis 35: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 40]; Test type: Superiority or Other; p = 0.68, mid-p exact binomial method
Statistical Analysis 36: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 42]; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 37: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 43]; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 38: Comparison: 13vPnC; Urticaria: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.91, mid-p exact binomial method
Statistical Analysis 39: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 42]; Test type: Superiority or Other; p = 0.14, mid-p exact binomial method
Statistical Analysis 40: Comparison: 13vPnC; Viral syndrome: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.03, mid-p exact binomial method
Statistical Analysis 41: Comparison: 13vPnC; Weakness: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 42: Comparison: 13vPnC; Wheezing: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.25, mid-p exact binomial method

6. Primary Outcome: Relative Risk of Medically Attended Events Between 30-day Risk Window and 30-day Self-control Window: Dose 1 Inpatient and Emergency Department Combined
Description: Relative risk for given event = incidence rate (risk window) / incidence rate (self-control window). Relative risk in inpatient and emergency department health care setting for Dose 1 was assessed by comparing the overall incidence rates of reported events in both settings per 1000 person-months occurring within 30 days after Dose 1 (30-day risk window) with the self-control period occurring during the subsequent 30 days (30-day self-control window). Relative risk and exact 2-sided 90% CIs were reported. Medically attended events were documented retrospectively according to ICD-9 coding. Results were reported for events reported in either of the windows.
Time Frame: 30 days after Dose 1 (risk window for Dose 1), 30 days after risk window (post-dose self-control window for Dose 1)
Population: as for baseline characteristics
Measure: Number (90% Confidence Interval); unit: ratio
Arm/Group | 13vPnC
Number analyzed (Participants) | 53902
ratio
  Abnormal involuntary movements | 1.52 [0.44 to 5.74]
  Acute bronchiolitis due to RSV | 1.93 [1.19 to 3.17]
  Acute febrile mucocutaneous lymph node syndrome | 0.91 [0.05 to 17.29]
  Acute otitis media | 0.70 [0.41 to 1.20]
  Acute pyelonephritis without RMN lesion | 1.14 [0.36 to 3.71]
  Adverse drug reaction | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Alkalosis | NA [1.95 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Apnea | 2.37 [1.01 to 6.03]
  Apparent life threatening event infant | 2.43 [1.12 to 5.63]
  Asthma with acute exacerbation | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Asthma, unspecified, unspecified status | 0.53 [0.23 to 1.16]
  Bronchiolitis | 0.77 [0.56 to 1.06]
  Bronchitis | 1.82 [0.21 to 26.39]
  Bronchospasm | 0.61 [0.24 to 1.46]
  Candidiasis of mouth | 4.10 [1.20 to 18.93]
  Cellulitis and abscess of trunk | 2.73 [0.41 to 35.48]
  Constipation | 0.63 [0.30 to 1.29]
  Croup | 0.58 [0.32 to 1.02]
  Dehydration | 1.00 [0.60 to 1.68]
  Dermatitis | 0.28 [0.11 to 0.65]
  Dyspnea | 1.58 [0.93 to 2.73]
  Failure to thrive | 1.72 [0.88 to 3.49]
  Fever | 1.39 [1.13 to 1.73]
  Fussy infant | 1.21 [0.83 to 1.78]
  Gastroenteritis | 0.57 [0.21 to 1.47]
  Hand, foot and mouth disease | NA [NA to 8.19] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Hematoma | 0.91 [0.05 to 17.29]
  Hypopotassemia | NA [0.42 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Lipoma of other specified sites | 0.46 [0.03 to 3.92]
  Methicillin susceptible Staphylococcus aureus | 4.55 [0.83 to 53.66]
  Nausea and vomiting | 0.69 [0.46 to 1.04]
  Neonatal bradycardia | NA [1.17 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Neonatal candida infection | 1.82 [0.21 to 26.39]
  Other diseases of nasal cavity and sinuses | 0.68 [0.43 to 1.06]
  Other specified cardiac dysrhythmias | 3.19 [0.88 to 15.19]
  Pilonidal cyst without mention of abscess | 2.36 [1.48 to 3.83]
  Pneumonia | 0.56 [0.34 to 0.92]
  Primary apnea of newborn | NA [1.56 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Rash | 1.02 [0.58 to 1.78]
  Respiratory syncytial virus | 2.73 [0.93 to 9.39]
  Retinopathy of prematurity stage 2 | NA [0.79 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Single seizure | 0.85 [0.44 to 1.61]
  Stridor | 0.73 [0.22 to 2.29]
  Subconjunctival hemorrhage | NA [0.42 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Umbilical hernia without obstruction/gangrene | 2.37 [1.01 to 6.03]
  Unspecified bacterial pneumonia | NA [1.17 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Unspecified septicemia | 3.03 [1.06 to 10.30]
  Urinary tract infection | 2.73 [1.56 to 4.97]
  Urticaria | 0.91 [0.21 to 3.90]
  Vaccines adverse reaction | NA [0.79 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Viral syndrome | 0.63 [0.42 to 0.93]
  Weakness | NA [0.42 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Wheezing | 0.55 [0.22 to 1.28]
Statistical Analysis 1: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.59, mid-p exact binomial method
Statistical Analysis 2: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.02, mid-p exact binomial method
Statistical Analysis 3: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.95, mid-p exact binomial method
Statistical Analysis 4: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p = 0.28, mid-p exact binomial method
Statistical Analysis 5: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.86, mid-p exact binomial method
Statistical Analysis 6: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 7: Comparison: 13vPnC; Alkalosis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.02, mid-p exact binomial method
Statistical Analysis 8: Comparison: 13vPnC; Apnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.10, mid-p exact binomial method
Statistical Analysis 9: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; p = 0.06, mid-p exact binomial method
Statistical Analysis 10: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 11: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; p = 0.19, mid-p exact binomial method
Statistical Analysis 12: Comparison: 13vPnC; Bronchiolitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.18, mid-p exact binomial method
Statistical Analysis 13: Comparison: 13vPnC; Bronchitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.68, mid-p exact binomial method
Statistical Analysis 14: Comparison: 13vPnC; Bronchospasm: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.35, mid-p exact binomial method
Statistical Analysis 15: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; p = 0.05, mid-p exact binomial method
Statistical Analysis 16: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 14]; Test type: Superiority or Other; p = 0.42, mid-p exact binomial method
Statistical Analysis 17: Comparison: 13vPnC; Constipation: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.29, mid-p exact binomial method
Statistical Analysis 18: Comparison: 13vPnC; Croup: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.11, mid-p exact binomial method
Statistical Analysis 19: Comparison: 13vPnC; Dehydration: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 1.00, mid-p exact binomial method
Statistical Analysis 20: Comparison: 13vPnC; Dermatitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 21: Comparison: 13vPnC; Dyspnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.16, mid-p exact binomial method
Statistical Analysis 22: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 20]; Test type: Superiority or Other; p = 0.19, mid-p exact binomial method
Statistical Analysis 23: Comparison: 13vPnC; Fever: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 24: Comparison: 13vPnC; Fussy infant: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.40, mid-p exact binomial method
Statistical Analysis 25: Comparison: 13vPnC; Gastroenteritis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.33, mid-p exact binomial method
Statistical Analysis 26: Comparison: 13vPnC; [analysis description as in outcome 5, analysis 23]; Test type: Superiority or Other; p = 0.48, mid-p exact binomial method
Statistical Analysis 27: Comparison: 13vPnC; Hematoma: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.95, mid-p exact binomial method
Statistical Analysis 28: Comparison: 13vPnC; Hypopotassemia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.27, mid-p exact binomial method
Statistical Analysis 29: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 25]; Test type: Superiority or Other; p = 0.57, mid-p exact binomial method
Statistical Analysis 30: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 26]; Test type: Superiority or Other; p = 0.15, mid-p exact binomial method
Statistical Analysis 31: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 27]; Test type: Superiority or Other; p = 0.14, mid-p exact binomial method
Statistical Analysis 32: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 28]; Test type: Superiority or Other; p = 0.08, mid-p exact binomial method
Statistical Analysis 33: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 29]; Test type: Superiority or Other; p = 0.68, mid-p exact binomial method
Statistical Analysis 34: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 30]; Test type: Superiority or Other; p = 0.15, mid-p exact binomial method
Statistical Analysis 35: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 31]; Test type: Superiority or Other; p = 0.14, mid-p exact binomial method
Statistical Analysis 36: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 32]; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 37: Comparison: 13vPnC; Pneumonia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.06, mid-p exact binomial method
Statistical Analysis 38: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 34]; Test type: Superiority or Other; p = 0.04, mid-p exact binomial method
Statistical Analysis 39: Comparison: 13vPnC; Rash: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.96, mid-p exact binomial method
Statistical Analysis 40: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 36]; Test type: Superiority or Other; p = 0.13, mid-p exact binomial method
Statistical Analysis 41: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 37]; Test type: Superiority or Other; p = 0.14, mid-p exact binomial method
Statistical Analysis 42: Comparison: 13vPnC; Single seizure: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.67, mid-p exact binomial method
Statistical Analysis 43: Comparison: 13vPnC; Stridor: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.65, mid-p exact binomial method
Statistical Analysis 44: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 37]; Test type: Superiority or Other; p = 0.27, mid-p exact binomial method
Statistical Analysis 45: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 40]; Test type: Superiority or Other; p = 0.10, mid-p exact binomial method
Statistical Analysis 46: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 41]; Test type: Superiority or Other; p = 0.08, mid-p exact binomial method
Statistical Analysis 47: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 42]; Test type: Superiority or Other; p = 0.08, mid-p exact binomial method
Statistical Analysis 48: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 43]; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 49: Comparison: 13vPnC; Urticaria: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.91, mid-p exact binomial method
Statistical Analysis 50: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 42]; Test type: Superiority or Other; p = 0.14, mid-p exact binomial method
Statistical Analysis 51: Comparison: 13vPnC; Viral syndrome: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.05, mid-p exact binomial method
Statistical Analysis 52: Comparison: 13vPnC; Weakness: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.27, mid-p exact binomial method
Statistical Analysis 53: Comparison: 13vPnC; Wheezing: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.25, mid-p exact binomial method

7. Primary Outcome: Relative Risk of Medically Attended Events Between 30-day Risk Window and 30-day Self-control Window: Dose 2 Inpatient
Description: Relative risk for given event = incidence rate (risk window) / incidence rate (self-control window). Relative risk in inpatient health care setting for Dose 2 was assessed by comparing the incidence rate of reported events in inpatient setting per 1000 person-months occurring within 30 days after Dose 2 (30-day risk window) with the self-control period occurring during the subsequent 30 days (30-day self-control window). Relative risk and exact 2-sided 90% CIs were reported. Medically attended events were documented retrospectively according to ICD-9 coding. Results were reported for events reported in either of the windows.
Time Frame: 30 days after Dose 2 (risk window for Dose 2), 30 days after risk window (post-dose self-control window for Dose 2)
Population: Analysis population included participants who started vaccination with 13vPnC within the first 6 months of life, were members of KPNC and received at least 2 doses of 13vPnC vaccine during the study observation period.
Measure: Number (90% Confidence Interval); unit: ratio
Groups:
- 13vPnC: Participants enrolled in Kaiser Permanente Northern California (KPNC) health maintenance organization who received 2 primary doses of 13-valent pneumococcal conjugate vaccine (13vPnC, Prevnar 13 or Prevenar 13) within the first 6 months of life at approximately 2, 4 months of age, according to the Advisory Committee on Immunization Practices (ACIP)-recommended schedule.
Arm/Group | 13vPnC
Number analyzed (Participants) | 49230
ratio
  Abnormal involuntary movements | 4.65 [0.84 to 54.82]
  Acute bronchiolitis due to RSV | 1.06 [0.58 to 1.96]
  Acute febrile mucocutaneous lymph node syndrome | 0.93 [0.05 to 17.67]
  Acute otitis media | 0.53 [0.17 to 1.51]
  Acute pyelonephritis without RMN lesion | NA [0.43 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Alkalosis | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Apnea | NA [NA to 2.01] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Apparent life threatening event infant | 0.23 [0.02 to 1.38]
  Asthma with acute exacerbation | 0.93 [0.05 to 17.67]
  Asthma, unspecified, unspecified status | 0.70 [0.18 to 2.60]
  Bronchiolitis | 1.63 [0.78 to 3.49]
  Bronchitis | 0.93 [0.05 to 17.67]
  Bronchospasm | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Cellulitis and abscess of trunk | 0.93 [0.05 to 17.67]
  Constipation | 2.79 [0.42 to 36.25]
  Croup | 1.24 [0.33 to 4.92]
  Dehydration | 1.01 [0.50 to 2.05]
  Dermatitis | 1.86 [0.43 to 9.78]
  Dyspnea | 0.93 [0.27 to 3.20]
  Failure to thrive | 1.16 [0.53 to 2.61]
  Fever | 0.93 [0.31 to 2.77]
  Fussy infant | NA [NA to 2.01] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Gastroenteritis | 0.93 [0.15 to 5.94]
  Hypopotassemia | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Lipoma of other specified sites | NA [0.43 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Methicillin susceptible Staphylococcus aureus | NA [0.81 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Nausea and vomiting | NA [NA to 8.37] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Other diseases of nasal cavity and sinuses | 0.31 [0.02 to 2.08]
  Other specified cardiac dysrhythmias | 2.79 [0.42 to 36.25]
  Pilonidal cyst without mention of abscess | 2.07 [1.08 to 4.13]
  Pneumonia | 0.78 [0.27 to 2.17]
  Primary apnea of newborn | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Rash | NA [NA to 8.37] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Retinopathy of prematurity stage 2 | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Single seizure | 0.47 [0.09 to 1.99]
  Stridor | 3.72 [0.63 to 45.53]
  Umbilical hernia without obstruction/gangrene | 3.72 [0.63 to 45.53]
  Unspecified bacterial pneumonia | 0.93 [0.05 to 17.67]
  Unspecified septicemia | 0.93 [0.05 to 17.67]
  Urinary tract infection | 0.66 [0.24 to 1.78]
  Urticaria | NA [NA to 8.37] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Viral syndrome | 1.24 [0.33 to 4.92]
  Weakness | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
Statistical Analysis 1: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.15, mid-p exact binomial method
Statistical Analysis 2: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.87, mid-p exact binomial method
Statistical Analysis 3: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.96, mid-p exact binomial method
Statistical Analysis 4: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p = 0.33, mid-p exact binomial method
Statistical Analysis 5: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.27, mid-p exact binomial method
Statistical Analysis 6: Comparison: 13vPnC; Alkalosis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 7: Comparison: 13vPnC; Apnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.23, mid-p exact binomial method
Statistical Analysis 8: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; p = 0.19, mid-p exact binomial method
Statistical Analysis 9: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.96, mid-p exact binomial method
Statistical Analysis 10: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; p = 0.66, mid-p exact binomial method
Statistical Analysis 11: Comparison: 13vPnC; Bronchiolitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.28, mid-p exact binomial method
Statistical Analysis 12: Comparison: 13vPnC; Bronchitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.96, mid-p exact binomial method
Statistical Analysis 13: Comparison: 13vPnC; Bronchospasm: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 14: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 14]; Test type: Superiority or Other; p = 0.96, mid-p exact binomial method
Statistical Analysis 15: Comparison: 13vPnC; Constipation: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.41, mid-p exact binomial method
Statistical Analysis 16: Comparison: 13vPnC; Croup: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.80, mid-p exact binomial method
Statistical Analysis 17: Comparison: 13vPnC; Dehydration: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.98, mid-p exact binomial method
Statistical Analysis 18: Comparison: 13vPnC; Dermatitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.51, mid-p exact binomial method
Statistical Analysis 19: Comparison: 13vPnC; Dyspnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.92, mid-p exact binomial method
Statistical Analysis 20: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 20]; Test type: Superiority or Other; p = 0.76, mid-p exact binomial method
Statistical Analysis 21: Comparison: 13vPnC; Fever: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.91, mid-p exact binomial method
Statistical Analysis 22: Comparison: 13vPnC; Fussy infant: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.23, mid-p exact binomial method
Statistical Analysis 23: Comparison: 13vPnC; Gastroenteritis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.95, mid-p exact binomial method
Statistical Analysis 24: Comparison: 13vPnC; Hypopotassemia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 25: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 25]; Test type: Superiority or Other; p = 0.27, mid-p exact binomial method
Statistical Analysis 26: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 26]; Test type: Superiority or Other; p = 0.14, mid-p exact binomial method
Statistical Analysis 27: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 27]; Test type: Superiority or Other; p = 0.48, mid-p exact binomial method
Statistical Analysis 28: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 30]; Test type: Superiority or Other; p = 0.34, mid-p exact binomial method
Statistical Analysis 29: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 31]; Test type: Superiority or Other; p = 0.41, mid-p exact binomial method
Statistical Analysis 30: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 32]; Test type: Superiority or Other; p = 0.07, mid-p exact binomial method
Statistical Analysis 31: Comparison: 13vPnC; Pneumonia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.69, mid-p exact binomial method
Statistical Analysis 32: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 34]; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 33: Comparison: 13vPnC; Rash: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.48, mid-p exact binomial method
Statistical Analysis 34: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 37]; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 35: Comparison: 13vPnC; Single seizure: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.40, mid-p exact binomial method
Statistical Analysis 36: Comparison: 13vPnC; Stridor: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.25, mid-p exact binomial method
Statistical Analysis 37: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 40]; Test type: Superiority or Other; p = 0.25, mid-p exact binomial method
Statistical Analysis 38: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 41]; Test type: Superiority or Other; p = 0.96, mid-p exact binomial method
Statistical Analysis 39: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 42]; Test type: Superiority or Other; p = 0.96, mid-p exact binomial method
Statistical Analysis 40: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 43]; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 41: Comparison: 13vPnC; Urticaria: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.48, mid-p exact binomial method
Statistical Analysis 42: Comparison: 13vPnC; Viral syndrome: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.80, mid-p exact binomial method
Statistical Analysis 43: Comparison: 13vPnC; Weakness: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method

8. Primary Outcome: Relative Risk of Medically Attended Events Between 30-day Risk Window and 30-day Self-control Window: Dose 2 Emergency Department
Description: Relative risk for given event = incidence rate (risk window) / incidence rate (self-control window). Relative risk in emergency department health care setting for Dose 2 was assessed by comparing the incidence rate of reported events in emergency department setting per 1000 person-months occurring within 30 days after Dose 2 (30-day risk window) with the self-control period occurring during the subsequent 30 days (30-day self-control window). Relative risk and exact 2-sided 90% CIs were reported. Medically attended events were documented retrospectively according to ICD-9 coding. Results were reported for events reported in either of the windows.
Time Frame: 30 days after Dose 2 (risk window for Dose 2), 30 days after risk window (post-dose self-control window for Dose 2)
Population: as for outcome 7
Measure: Number (90% Confidence Interval); unit: ratio
Arm/Group | 13vPnC
Number analyzed (Participants) | 49230
ratio
  Abnormal involuntary movements | NA [0.43 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Acute bronchiolitis due to RSV | 2.79 [1.21 to 7.00]
  Acute otitis media | 0.57 [0.39 to 0.82]
  Adverse drug reaction | 0.93 [0.15 to 5.94]
  Apnea | NA [NA to 2.01] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Apparent life threatening event infant | 0.31 [0.02 to 2.08]
  Asthma with acute exacerbation | NA [NA to 8.37] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Asthma, unspecified, unspecified status | 0.93 [0.45 to 1.90]
  Bronchiolitis | 0.84 [0.62 to 1.14]
  Bronchitis | 1.16 [0.37 to 3.79]
  Bronchospasm | 1.24 [0.60 to 2.63]
  Candidiasis of mouth | 0.93 [0.15 to 5.94]
  Constipation | 0.68 [0.31 to 1.47]
  Croup | 0.87 [0.60 to 1.24]
  Dehydration | 1.03 [0.48 to 2.25]
  Dermatitis | 0.47 [0.19 to 1.06]
  Dyspnea | 0.84 [0.38 to 1.81]
  Failure to thrive | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Fever | 1.15 [0.94 to 1.40]
  Fussy infant | 1.49 [0.77 to 2.96]
  Gastroenteritis | 1.05 [0.59 to 1.86]
  Hand, foot and mouth disease | 1.86 [0.22 to 26.96]
  Hematoma | NA [NA to 8.37] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Nausea and vomiting | 0.70 [0.51 to 0.97]
  Neonatal candida infection | NA [0.43 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Other diseases of nasal cavity and sinuses | 2.92 [1.45 to 6.25]
  Pneumonia | 0.72 [0.44 to 1.17]
  Rash | 0.73 [0.41 to 1.30]
  Respiratory syncytial virus | 0.31 [0.02 to 2.08]
  Single seizure | 1.40 [0.58 to 3.48]
  Stomatitis | NA [NA to 8.37] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Stridor | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Subconjunctival hemorrhage | NA [0.43 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Umbilical hernia without obstruction/gangrene | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Unspecified septicemia | NA [NA to 8.37] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Urinary tract infection | 1.20 [0.71 to 2.07]
  Urticaria | 0.83 [0.36 to 1.87]
  Vaccines adverse reaction | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Viral syndrome | 0.59 [0.39 to 0.88]
  Weakness | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Wheezing | 0.80 [0.47 to 1.36]
Statistical Analysis 1: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.27, mid-p exact binomial method
Statistical Analysis 2: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.04, mid-p exact binomial method
Statistical Analysis 3: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p = 0.01, mid-p exact binomial method
Statistical Analysis 4: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.95, mid-p exact binomial method
Statistical Analysis 5: Comparison: 13vPnC; Apnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.23, mid-p exact binomial method
Statistical Analysis 6: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; p = 0.34, mid-p exact binomial method
Statistical Analysis 7: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.48, mid-p exact binomial method
Statistical Analysis 8: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; p = 0.87, mid-p exact binomial method
Statistical Analysis 9: Comparison: 13vPnC; Bronchiolitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.35, mid-p exact binomial method
Statistical Analysis 10: Comparison: 13vPnC; Bronchitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.84, mid-p exact binomial method
Statistical Analysis 11: Comparison: 13vPnC; Bronchospasm: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.64, mid-p exact binomial method
Statistical Analysis 12: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; p = 0.95, mid-p exact binomial method
Statistical Analysis 13: Comparison: 13vPnC; Constipation: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.41, mid-p exact binomial method
Statistical Analysis 14: Comparison: 13vPnC; Croup: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.51, mid-p exact binomial method
Statistical Analysis 15: Comparison: 13vPnC; Dehydration: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.95, mid-p exact binomial method
Statistical Analysis 16: Comparison: 13vPnC; Dermatitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.13, mid-p exact binomial method
Statistical Analysis 17: Comparison: 13vPnC; Dyspnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.70, mid-p exact binomial method
Statistical Analysis 18: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 20]; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 19: Comparison: 13vPnC; Fever: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.25, mid-p exact binomial method
Statistical Analysis 20: Comparison: 13vPnC; Fussy infant: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.33, mid-p exact binomial method
Statistical Analysis 21: Comparison: 13vPnC; Gastroenteritis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.90, mid-p exact binomial method
Statistical Analysis 22: Comparison: 13vPnC; [analysis description as in outcome 5, analysis 23]; Test type: Superiority or Other; p = 0.67, mid-p exact binomial method
Statistical Analysis 23: Comparison: 13vPnC; Hematoma: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.48, mid-p exact binomial method
Statistical Analysis 24: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 27]; Test type: Superiority or Other; p = 0.07, mid-p exact binomial method
Statistical Analysis 25: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 29]; Test type: Superiority or Other; p = 0.27, mid-p exact binomial method
Statistical Analysis 26: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 30]; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 27: Comparison: 13vPnC; Pneumonia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.27, mid-p exact binomial method
Statistical Analysis 28: Comparison: 13vPnC; Rash: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.38, mid-p exact binomial method
Statistical Analysis 29: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 36]; Test type: Superiority or Other; p = 0.34, mid-p exact binomial method
Statistical Analysis 30: Comparison: 13vPnC; Single seizure: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.54, mid-p exact binomial method
Statistical Analysis 31: Comparison: 13vPnC; Stomatitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.48, mid-p exact binomial method
Statistical Analysis 32: Comparison: 13vPnC; Stridor: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 33: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 37]; Test type: Superiority or Other; p = 0.27, mid-p exact binomial method
Statistical Analysis 34: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 40]; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 35: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 42]; Test type: Superiority or Other; p = 0.48, mid-p exact binomial method
Statistical Analysis 36: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 43]; Test type: Superiority or Other; p = 0.57, mid-p exact binomial method
Statistical Analysis 37: Comparison: 13vPnC; Urticaria: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.70, mid-p exact binomial method
Statistical Analysis 38: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 42]; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 39: Comparison: 13vPnC; Viral syndrome: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.03, mid-p exact binomial method
Statistical Analysis 40: Comparison: 13vPnC; Weakness: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 41: Comparison: 13vPnC; Wheezing: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.48, mid-p exact binomial method

9. Primary Outcome: Relative Risk of Medically Attended Events Between 30-day Risk Window and 30-day Self-control Window: Dose 2 Inpatient and Emergency Department Combined
Description: Relative risk for given event = incidence rate (risk window) / incidence rate (self-control window). Relative risk in inpatient and emergency department health care setting for Dose 2 was assessed by comparing the overall incidence rates of reported events in both settings per 1000 person-months occurring within 30 days after Dose 2 (30-day risk window) with the self-control period occurring during the subsequent 30 days (30-day self-control window). Relative risk and exact 2-sided 90% CIs were reported. Medically attended events were documented retrospectively according to ICD-9 coding. Results reported for events reported in either of the windows.
Time Frame: 30 days after Dose 2 (risk window for Dose 2), 30 days after risk window (post-dose self-control window for Dose 2)
Population: as for outcome 7
Measure: Number (90% Confidence Interval); unit: ratio
Arm/Group | 13vPnC
Number analyzed (Participants) | 49230
ratio
  Abnormal involuntary movements | 6.51 [1.29 to 73.39]
  Acute bronchiolitis due to RSV | 1.45 [0.88 to 2.40]
  Acute febrile mucocutaneous lymph node syndrome | 0.93 [0.05 to 17.67]
  Acute otitis media | 0.55 [0.38 to 0.79]
  Acute pyelonephritis without RMN lesion | NA [0.43 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Adverse drug reaction | 0.93 [0.15 to 5.94]
  Alkalosis | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Apnea | NA [NA to 0.72] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Apparent life threatening event infant | 0.31 [0.06 to 1.16]
  Asthma with acute exacerbation | 0.47 [0.03 to 4.00]
  Asthma, unspecified, unspecified status | 0.81 [0.43 to 1.51]
  Bronchiolitis | 0.86 [0.65 to 1.15]
  Bronchitis | 1.12 [0.40 to 3.20]
  Bronchospasm | 1.34 [0.65 to 2.82]
  Candidiasis of mouth | 0.93 [0.15 to 5.94]
  Cellulitis and abscess of trunk | 0.93 [0.05 to 17.67]
  Constipation | 0.85 [0.42 to 1.71]
  Croup | 0.87 [0.61 to 1.23]
  Dehydration | 0.78 [0.44 to 1.37]
  Dermatitis | 0.64 [0.31 to 1.32]
  Dyspnea | 0.86 [0.45 to 1.64]
  Failure to thrive | 1.16 [0.53 to 2.61]
  Fever | 1.13 [0.93 to 1.38]
  Fussy infant | 1.24 [0.66 to 2.37]
  Gastroenteritis | 1.03 [0.60 to 1.78]
  Hand, foot and mouth disease | 1.86 [0.22 to 26.96]
  Hematoma | NA [NA to 8.37] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Hypopotassemia | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Lipoma of other specified sites | NA [0.43 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Methicillin susceptible Staphylococcus aureus | NA [0.81 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Nausea and vomiting | 0.70 [0.51 to 0.97]
  Neonatal candida infection | NA [0.43 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Other diseases of nasal cavity and sinuses | 2.14 [1.16 to 4.10]
  Other specified cardiac dysrhythmias | 2.79 [0.42 to 36.25]
  Pilonidal cyst without mention of abscess | 2.07 [1.08 to 4.13]
  Pneumonia | 0.77 [0.49 to 1.21]
  Primary apnea of newborn | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Rash | 0.70 [0.39 to 1.23]
  Respiratory syncytial virus | 0.31 [0.02 to 2.08]
  Retinopathy of prematurity stage 2 | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Single seizure | 0.84 [0.38 to 1.81]
  Stomatitis | NA [NA to 8.37] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Stridor | 3.72 [0.63 to 45.53]
  Subconjunctival hemorrhage | NA [0.43 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Umbilical hernia without obstruction/gangrene | 4.65 [0.84 to 54.82]
  Unspecified bacterial pneumonia | 0.93 [0.05 to 17.67]
  Unspecified septicemia | 0.93 [0.05 to 17.67]
  Urinary tract infection | 1.09 [0.68 to 1.75]
  Urticaria | 0.74 [0.33 to 1.64]
  Vaccines adverse reaction | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Viral syndrome | 0.61 [0.42 to 0.90]
  Weakness | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Wheezing | 0.80 [0.47 to 1.36]
Statistical Analysis 1: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.05, mid-p exact binomial method
Statistical Analysis 2: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.22, mid-p exact binomial method
Statistical Analysis 3: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.96, mid-p exact binomial method
Statistical Analysis 4: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 5: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.27, mid-p exact binomial method
Statistical Analysis 6: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.95, mid-p exact binomial method
Statistical Analysis 7: Comparison: 13vPnC; Alkalosis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 8: Comparison: 13vPnC; Apnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.05, mid-p exact binomial method
Statistical Analysis 9: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; p = 0.15, mid-p exact binomial method
Statistical Analysis 10: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.58, mid-p exact binomial method
Statistical Analysis 11: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; p = 0.57, mid-p exact binomial method
Statistical Analysis 12: Comparison: 13vPnC; Bronchiolitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.39, mid-p exact binomial method
Statistical Analysis 13: Comparison: 13vPnC; Bronchitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.87, mid-p exact binomial method
Statistical Analysis 14: Comparison: 13vPnC; Bronchospasm: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.51, mid-p exact binomial method
Statistical Analysis 15: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; p = 0.95, mid-p exact binomial method
Statistical Analysis 16: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 14]; Test type: Superiority or Other; p = 0.96, mid-p exact binomial method
Statistical Analysis 17: Comparison: 13vPnC; Constipation: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.71, mid-p exact binomial method
Statistical Analysis 18: Comparison: 13vPnC; Croup: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.51, mid-p exact binomial method
Statistical Analysis 19: Comparison: 13vPnC; Dehydration: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.48, mid-p exact binomial method
Statistical Analysis 20: Comparison: 13vPnC; Dermatitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.32, mid-p exact binomial method
Statistical Analysis 21: Comparison: 13vPnC; Dyspnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.71, mid-p exact binomial method
Statistical Analysis 22: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 20]; Test type: Superiority or Other; p = 0.76, mid-p exact binomial method
Statistical Analysis 23: Comparison: 13vPnC; Fever: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.29, mid-p exact binomial method
Statistical Analysis 24: Comparison: 13vPnC; Fussy infant: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.58, mid-p exact binomial method
Statistical Analysis 25: Comparison: 13vPnC; Gastroenteritis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.92, mid-p exact binomial method
Statistical Analysis 26: Comparison: 13vPnC; [analysis description as in outcome 5, analysis 23]; Test type: Superiority or Other; p = 0.67, mid-p exact binomial method
Statistical Analysis 27: Comparison: 13vPnC; Hematoma: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.48, mid-p exact binomial method
Statistical Analysis 28: Comparison: 13vPnC; Hypopotassemia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 29: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 25]; Test type: Superiority or Other; p = 0.27, mid-p exact binomial method
Statistical Analysis 30: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 26]; Test type: Superiority or Other; p = 0.14, mid-p exact binomial method
Statistical Analysis 31: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 27]; Test type: Superiority or Other; p = 0.07, mid-p exact binomial method
Statistical Analysis 32: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 29]; Test type: Superiority or Other; p = 0.27, mid-p exact binomial method
Statistical Analysis 33: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 30]; Test type: Superiority or Other; p = 0.04, mid-p exact binomial method
Statistical Analysis 34: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 31]; Test type: Superiority or Other; p = 0.41, mid-p exact binomial method
Statistical Analysis 35: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 32]; Test type: Superiority or Other; p = 0.07, mid-p exact binomial method
Statistical Analysis 36: Comparison: 13vPnC; Pneumonia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.35, mid-p exact binomial method
Statistical Analysis 37: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 34]; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 38: Comparison: 13vPnC; Rash: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.30, mid-p exact binomial method
Statistical Analysis 39: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 36]; Test type: Superiority or Other; p = 0.34, mid-p exact binomial method
Statistical Analysis 40: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 37]; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 41: Comparison: 13vPnC; Single seizure: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.70, mid-p exact binomial method
Statistical Analysis 42: Comparison: 13vPnC; Stomatitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.48, mid-p exact binomial method
Statistical Analysis 43: Comparison: 13vPnC; Stridor: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.25, mid-p exact binomial method
Statistical Analysis 44: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 37]; Test type: Superiority or Other; p = 0.27, mid-p exact binomial method
Statistical Analysis 45: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 40]; Test type: Superiority or Other; p = 0.15, mid-p exact binomial method
Statistical Analysis 46: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 41]; Test type: Superiority or Other; p = 0.96, mid-p exact binomial method
Statistical Analysis 47: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 42]; Test type: Superiority or Other; p = 0.96, mid-p exact binomial method
Statistical Analysis 48: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 43]; Test type: Superiority or Other; p = 0.76, mid-p exact binomial method
Statistical Analysis 49: Comparison: 13vPnC; Urticaria: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.54, mid-p exact binomial method
Statistical Analysis 50: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 42]; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 51: Comparison: 13vPnC; Viral syndrome: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.03, mid-p exact binomial method
Statistical Analysis 52: Comparison: 13vPnC; Weakness: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 53: Comparison: 13vPnC; Wheezing: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.48, mid-p exact binomial method

10. Primary Outcome: Relative Risk of Medically Attended Events Between 30-day Risk Window and 30-day Self-control Window: Dose 3 Inpatient
Description: Relative risk for given event = incidence rate (risk window) / incidence rate (self-control window). Relative risk in inpatient health care setting for Dose 3 was assessed by comparing the incidence rate of reported events in inpatient setting per 1000 person-months occurring within 30 days after Dose 3 (30-day risk window) with the self-control period occurring during the subsequent 30 days (30-day self-control window). Relative risk and exact 2-sided 90% CIs were reported. Medically attended events were documented retrospectively according to ICD-9 coding. Results were reported for events reported in either of the windows.
Time Frame: 30 days after Dose 3 (risk window for Dose 3), 30 days after risk window (post-dose self-control window for Dose 3)
Population: Analysis population included participants who started vaccination with 13vPnC within the first 6 months of life, were members of KPNC and received at least 3 doses of 13vPnC vaccine during the study observation period.
Measure: Number (90% Confidence Interval); unit: ratio
Arm/Group | 13vPnC
Number analyzed (Participants) | 44178
ratio
  Abnormal involuntary movements | 1.97 [0.23 to 28.51]
  Acute bronchiolitis due to RSV | 1.15 [0.60 to 2.23]
  Acute febrile mucocutaneous lymph node syndrome | NA [1.68 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Acute otitis media | 1.38 [0.51 to 3.83]
  Acute pyelonephritis without RMN lesion | 2.95 [0.44 to 38.33]
  Alkalosis | NA [NA to 8.85] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Apnea | 0.98 [0.05 to 18.69]
  Apparent life threatening event infant | NA [0.85 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Asthma with acute exacerbation | NA [0.45 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Asthma, unspecified, unspecified status | 0.39 [0.14 to 1.03]
  Bronchiolitis | 1.35 [0.62 to 3.00]
  Bronchitis | NA [NA to 8.85] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Candidiasis of mouth | 1.97 [0.23 to 28.51]
  Cellulitis and abscess of trunk | NA [NA to 2.13] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Constipation | 0.66 [0.21 to 1.94]
  Croup | 1.48 [0.30 to 8.32]
  Dehydration | 1.35 [0.79 to 2.35]
  Dermatitis | 0.98 [0.29 to 3.38]
  Dyspnea | 0.14 [0.01 to 0.71]
  Failure to thrive | 1.15 [0.45 to 2.99]
  Fever | 0.82 [0.29 to 2.29]
  Fussy infant | 0.98 [0.05 to 18.69]
  Gastroenteritis | NA [0.85 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Hand, foot and mouth disease | NA [0.11 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Hypopotassemia | NA [0.45 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Lipoma of other specified sites | 0.33 [0.03 to 2.20]
  Methicillin susceptible Staphylococcus aureus | 0.20 [0.02 to 1.08]
  Nausea and vomiting | NA [0.11 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Other diseases of nasal cavity and sinuses | 0.98 [0.05 to 18.69]
  Other specified cardiac dysrhythmias | 1.97 [0.23 to 28.51]
  Pilonidal cyst without mention of abscess | 0.86 [0.36 to 2.06]
  Pneumonia | 1.11 [0.49 to 2.53]
  Rash | 0.49 [0.09 to 2.11]
  Respiratory syncytial virus | NA [NA to 8.85] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Single seizure | 0.61 [0.23 to 1.59]
  Stridor | 0.98 [0.05 to 18.69]
  Subconjunctival hemorrhage | NA [NA to 8.85] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Umbilical hernia without obstruction/gangrene | 1.97 [0.23 to 28.51]
  Unspecified bacterial pneumonia | 0.98 [0.05 to 18.69]
  Unspecified septicemia | NA [NA to 8.85] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Urinary tract infection | 0.39 [0.08 to 1.56]
  Viral syndrome | 0.25 [0.02 to 1.46]
  Wheezing | 0.98 [0.23 to 4.21]
Statistical Analysis 1: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0 .63, mid-p exact binomial method
Statistical Analysis 2: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.73, mid-p exact binomial method
Statistical Analysis 3: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.03, mid-p exact binomial method
Statistical Analysis 4: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p = 0.60, mid-p exact binomial method
Statistical Analysis 5: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.38, mid-p exact binomial method
Statistical Analysis 6: Comparison: 13vPnC; Alkalosis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 7: Comparison: 13vPnC; Apnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.99, mid-p exact binomial method
Statistical Analysis 8: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; p = 0.13, mid-p exact binomial method
Statistical Analysis 9: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.25, mid-p exact binomial method
Statistical Analysis 10: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; p = 0.11, mid-p exact binomial method
Statistical Analysis 11: Comparison: 13vPnC; Bronchiolitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.53, mid-p exact binomial method
Statistical Analysis 12: Comparison: 13vPnC; Bronchitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 13: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; p = 0.63, mid-p exact binomial method
Statistical Analysis 14: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 14]; Test type: Superiority or Other; p = 0.25, mid-p exact binomial method
Statistical Analysis 15: Comparison: 13vPnC; Constipation: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.53, mid-p exact binomial method
Statistical Analysis 16: Comparison: 13vPnC; Croup: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.70, mid-p exact binomial method
Statistical Analysis 17: Comparison: 13vPnC; Dehydration: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.36, mid-p exact binomial method
Statistical Analysis 18: Comparison: 13vPnC; Dermatitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.98, mid-p exact binomial method
Statistical Analysis 19: Comparison: 13vPnC; Dyspnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.04, mid-p exact binomial method
Statistical Analysis 20: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 20]; Test type: Superiority or Other; p = 0.81, mid-p exact binomial method
Statistical Analysis 21: Comparison: 13vPnC; Fever: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.75, mid-p exact binomial method
Statistical Analysis 22: Comparison: 13vPnC; Fussy infant: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.99, mid-p exact binomial method
Statistical Analysis 23: Comparison: 13vPnC; Gastroenteritis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.13, mid-p exact binomial method
Statistical Analysis 24: Comparison: 13vPnC; [analysis description as in outcome 5, analysis 23]; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 25: Comparison: 13vPnC; Hypopotassemia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.25, mid-p exact binomial method
Statistical Analysis 26: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 25]; Test type: Superiority or Other; p = 0.37, mid-p exact binomial method
Statistical Analysis 27: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 26]; Test type: Superiority or Other; p = 0.12, mid-p exact binomial method
Statistical Analysis 28: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 27]; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 29: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 30]; Test type: Superiority or Other; p = 0.99, mid-p exact binomial method
Statistical Analysis 30: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 31]; Test type: Superiority or Other; p = 0.63, mid-p exact binomial method
Statistical Analysis 31: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 32]; Test type: Superiority or Other; p = 0.78, mid-p exact binomial method
Statistical Analysis 32: Comparison: 13vPnC; Pneumonia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.84, mid-p exact binomial method
Statistical Analysis 33: Comparison: 13vPnC; Rash: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.44, mid-p exact binomial method
Statistical Analysis 34: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 36]; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 35: Comparison: 13vPnC; Single seizure: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.41, mid-p exact binomial method
Statistical Analysis 36: Comparison: 13vPnC; Stridor: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.99, mid-p exact binomial method
Statistical Analysis 37: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 37]; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 38: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 40]; Test type: Superiority or Other; p = 0.63, mid-p exact binomial method
Statistical Analysis 39: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 41]; Test type: Superiority or Other; p = 0.99, mid-p exact binomial method
Statistical Analysis 40: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 42]; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 41: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 43]; Test type: Superiority or Other; p = 0.28, mid-p exact binomial method
Statistical Analysis 42: Comparison: 13vPnC; Viral syndrome: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.21, mid-p exact binomial method
Statistical Analysis 43: Comparison: 13vPnC; Wheezing: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.98, mid-p exact binomial method

11. Primary Outcome: Relative Risk of Medically Attended Events Between 30-day Risk Window and 30-day Self-control Window: Dose 3 Emergency Department
Description: Relative risk for given event = incidence rate (risk window) / incidence rate (self-control window). Relative risk in emergency department health care setting for Dose 3 was assessed by comparing the incidence rate of reported events in emergency department setting per 1000 person-months occurring within 30 days after Dose 3 (30-day risk window) with the self-control period occurring during the subsequent 30 days (30-day self-control window). Relative risk and its corresponding exact 2-sided 90% confidence CIs were reported. Medically attended events were documented retrospectively according to ICD-9 coding. Results were reported for events reported in either of the windows.
Time Frame: 30 days after Dose 3 (risk window for Dose 3), 30 days after risk window (post-dose self-control window for Dose 3)
Population: as for outcome 10
Measure: Number (90% Confidence Interval); unit: ratio
Arm/Group | 13vPnC
Number analyzed (Participants) | 44178
ratio
  Abnormal involuntary movements | NA [0.11 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Acute bronchiolitis due to RSV | 0.84 [0.32 to 2.16]
  Acute febrile mucocutaneous lymph node syndrome | NA [NA to 8.85] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Acute otitis media | 0.90 [0.68 to 1.19]
  Acute pyelonephritis without RMN lesion | NA [0.11 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Adverse drug reaction | 0.49 [0.03 to 4.23]
  Apnea | NA [0.11 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Apparent life threatening event infant | NA [0.11 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Asthma with acute exacerbation | NA [0.45 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Asthma, unspecified, unspecified status | 0.74 [0.39 to 1.39]
  Bronchiolitis | 1.29 [0.92 to 1.81]
  Bronchitis | 0.42 [0.12 to 1.31]
  Bronchospasm | 1.97 [0.92 to 4.39]
  Candidiasis of mouth | 0.25 [0.02 to 1.46]
  Cellulitis and abscess of trunk | NA [NA to 8.85] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Constipation | 1.09 [0.51 to 2.38]
  Croup | 1.26 [0.89 to 1.80]
  Dehydration | 1.12 [0.69 to 1.85]
  Dermatitis | 1.97 [0.72 to 5.89]
  Dyspnea | 2.62 [0.87 to 9.16]
  Failure to thrive | 0.98 [0.05 to 18.69]
  Fever | 1.07 [0.90 to 1.28]
  Fussy infant | 0.84 [0.43 to 1.62]
  Gastroenteritis | 0.51 [0.28 to 0.92]
  Hand, foot and mouth disease | 1.31 [0.35 to 5.21]
  Hematoma | 0.98 [0.15 to 6.28]
  Nausea and vomiting | 1.12 [0.85 to 1.50]
  Neonatal candida infection | NA [0.45 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Other diseases of nasal cavity and sinuses | 0.91 [0.48 to 1.74]
  Other specified cardiac dysrhythmias | NA [0.45 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Pneumonia | 1.14 [0.79 to 1.66]
  Rash | 0.66 [0.35 to 1.21]
  Respiratory syncytial virus | 0.49 [0.13 to 1.59]
  Single seizure | 1.15 [0.45 to 2.99]
  Stomatitis | NA [NA to 8.85] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Stridor | NA [1.26 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Umbilical hernia without obstruction/gangrene | NA [NA to 8.85] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Unspecified septicemia | NA [NA to 2.13] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Urinary tract infection | 1.18 [0.66 to 2.12]
  Urticaria | 0.98 [0.46 to 2.09]
  Viral syndrome | 0.81 [0.57 to 1.14]
  Weakness | NA [0.45 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Wheezing | 2.26 [1.22 to 4.34]
Statistical Analysis 1: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 2: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.77, mid-p exact binomial method
Statistical Analysis 3: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 4: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p = 0.55, mid-p exact binomial method
Statistical Analysis 5: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 6: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.62, mid-p exact binomial method
Statistical Analysis 7: Comparison: 13vPnC; Apnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 8: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 9: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.25, mid-p exact binomial method
Statistical Analysis 10: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; p = 0.43, mid-p exact binomial method
Statistical Analysis 11: Comparison: 13vPnC; Bronchiolitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.22, mid-p exact binomial method
Statistical Analysis 12: Comparison: 13vPnC; Bronchitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.22, mid-p exact binomial method
Statistical Analysis 13: Comparison: 13vPnC; Bronchospasm: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.14, mid-p exact binomial method
Statistical Analysis 14: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; p = 0.21, mid-p exact binomial method
Statistical Analysis 15: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 14]; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 16: Comparison: 13vPnC; Constipation: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.85, mid-p exact binomial method
Statistical Analysis 17: Comparison: 13vPnC; Croup: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.28, mid-p exact binomial method
Statistical Analysis 18: Comparison: 13vPnC; Dehydration: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.70, mid-p exact binomial method
Statistical Analysis 19: Comparison: 13vPnC; Dermatitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.28, mid-p exact binomial method
Statistical Analysis 20: Comparison: 13vPnC; Dyspnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.15, mid-p exact binomial method
Statistical Analysis 21: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 20]; Test type: Superiority or Other; p = 0.99, mid-p exact binomial method
Statistical Analysis 22: Comparison: 13vPnC; Fever: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.51, mid-p exact binomial method
Statistical Analysis 23: Comparison: 13vPnC; Fussy infant: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.67, mid-p exact binomial method
Statistical Analysis 24: Comparison: 13vPnC; Gastroenteritis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.06, mid-p exact binomial method
Statistical Analysis 25: Comparison: 13vPnC; [analysis description as in outcome 5, analysis 23]; Test type: Superiority or Other; p = 0.74, mid-p exact binomial method
Statistical Analysis 26: Comparison: 13vPnC; Hematoma: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.99, mid-p exact binomial method
Statistical Analysis 27: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 27]; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 28: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 29]; Test type: Superiority or Other; p = 0.25, mid-p exact binomial method
Statistical Analysis 29: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 30]; Test type: Superiority or Other; p = 0.82, mid-p exact binomial method
Statistical Analysis 30: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 31]; Test type: Superiority or Other; p = 0.25, mid-p exact binomial method
Statistical Analysis 31: Comparison: 13vPnC; Pneumonia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.55, mid-p exact binomial method
Statistical Analysis 32: Comparison: 13vPnC; Rash: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.26, mid-p exact binomial method
Statistical Analysis 33: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 36]; Test type: Superiority or Other; p = 0.33, mid-p exact binomial method
Statistical Analysis 34: Comparison: 13vPnC; Single seizure: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.81, mid-p exact binomial method
Statistical Analysis 35: Comparison: 13vPnC; Stomatitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 36: Comparison: 13vPnC; Stridor: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.06, mid-p exact binomial method
Statistical Analysis 37: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 40]; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 38: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 42]; Test type: Superiority or Other; p = 0.25, mid-p exact binomial method
Statistical Analysis 39: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 43]; Test type: Superiority or Other; p = 0.64, mid-p exact binomial method
Statistical Analysis 40: Comparison: 13vPnC; Urticaria: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.97, mid-p exact binomial method
Statistical Analysis 41: Comparison: 13vPnC; Viral syndrome: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.31, mid-p exact binomial method
Statistical Analysis 42: Comparison: 13vPnC; Weakness: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.25, mid-p exact binomial method
Statistical Analysis 43: Comparison: 13vPnC; Wheezing: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.03, mid-p exact binomial method

12. Primary Outcome: Relative Risk of Medically Attended Events Between 30-day Risk Window and 30-day Self-control Window: Dose 3 Inpatient and Emergency Department Combined
Description: Relative risk for given event=incidence rate(risk window)/incidence rate(self-control window). Relative risk in inpatient and emergency department health care setting for Dose 3 was assessed by comparing the overall incidence rates of reported events in both settings per 1000 person-months occurring within 30 days after Dose 3 (30-day risk window) with the self-control period occurring during the subsequent 30 days (30-day self-control window). Relative risk and exact 2-sided 90% CIs were reported. Medically attended events were documented retrospectively according to ICD-9 coding. Results reported for events reported in either of the windows.
Time Frame: 30 days after Dose 3 (risk window for Dose 3), 30 days after risk window (post-dose self-control window for Dose 3)
Population: as for outcome 10
Measure: Number (90% Confidence Interval); unit: ratio
Arm/Group | 13vPnC
Number analyzed (Participants) | 44178
ratio
  Abnormal involuntary movements | 2.95 [0.44 to 38.33]
  Acute bronchiolitis due to RSV | 1.10 [0.63 to 1.92]
  Acute febrile mucocutaneous lymph node syndrome | 4.92 [0.89 to 57.98]
  Acute otitis media | 0.95 [0.72 to 1.24]
  Acute pyelonephritis without RMN lesion | 3.93 [0.66 to 48.16]
  Adverse drug reaction | 0.49 [0.03 to 4.23]
  Alkalosis | NA [NA to 8.85] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Apnea | 0.98 [0.05 to 18.69]
  Apparent life threatening event infant | NA [0.85 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Asthma with acute exacerbation | NA [1.26 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Asthma, unspecified, unspecified status | 0.63 [0.37 to 1.07]
  Bronchiolitis | 1.33 [0.97 to 1.85]
  Bronchitis | 0.37 [0.11 to 1.11]
  Bronchospasm | 1.97 [0.92 to 4.39]
  Candidiasis of mouth | 0.39 [0.08 to 1.56]
  Cellulitis and abscess of trunk | NA [NA to 1.14] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Constipation | 0.85 [0.45 to 1.60]
  Croup | 1.29 [0.91 to 1.83]
  Dehydration | 1.13 [0.77 to 1.67]
  Dermatitis | 1.69 [0.77 to 3.84]
  Dyspnea | 0.79 [0.35 to 1.74]
  Failure to thrive | 1.31 [0.53 to 3.34]
  Fever | 1.05 [0.88 to 1.25]
  Fussy infant | 0.85 [0.45 to 1.60]
  Gastroenteritis | 0.64 [0.37 to 1.11]
  Hand, foot and mouth disease | 1.64 [0.48 to 6.20]
  Hematoma | 0.98 [0.15 to 6.28]
  Hypopotassemia | NA [0.45 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Lipoma of other specified sites | 0.33 [0.03 to 2.20]
  Methicillin susceptible Staphylococcus aureus | 0.20 [0.02 to 1.08]
  Nausea and vomiting | 1.12 [0.85 to 1.50]
  Neonatal candida infection | NA [0.45 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Other diseases of nasal cavity and sinuses | 0.92 [0.49 to 1.71]
  Other specified cardiac dysrhythmias | 2.95 [0.44 to 38.34]
  Pilonidal cyst without mention of abscess | 0.86 [0.36 to 2.06]
  Pneumonia | 1.10 [0.77 to 1.58]
  Rash | 0.63 [0.35 to 1.10]
  Respiratory syncytial virus | 0.42 [0.12 to 1.31]
  Single seizure | 0.91 [0.46 to 1.77]
  Stomatitis | NA [NA to 8.85] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Stridor | 4.92 [0.89 to 57.98]
  Subconjunctival hemorrhage | NA [NA to 8.85] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Umbilical hernia without obstruction/gangrene | 0.98 [0.15 to 6.28]
  Unspecified bacterial pneumonia | 0.98 [0.05 to 18.69]
  Unspecified septicemia | NA [NA to 2.13] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Urinary tract infection | 0.98 [0.58 to 1.66]
  Urticaria | 0.98 [0.46 to 2.09]
  Viral syndrome | 0.76 [0.54 to 1.07]
  Weakness | NA [0.45 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Wheezing | 2.13 [1.21 to 3.87]
Statistical Analysis 1: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.38, mid-p exact binomial method
Statistical Analysis 2: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.78, mid-p exact binomial method
Statistical Analysis 3: Comparison: 13vPnC; Acute febrile mucocutaneous lymph node syndrome: p-value was estimated using the mid-p exact binomial method.The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.13, mid-p exact binomial method
Statistical Analysis 4: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p = 0.73, mid-p exact binomial method
Statistical Analysis 5: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.23, mid-p exact binomial method
Statistical Analysis 6: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.62, mid-p exact binomial method
Statistical Analysis 7: Comparison: 13vPnC; Alkalosis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 8: Comparison: 13vPnC; Apnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.99, mid-p exact binomial method
Statistical Analysis 9: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; p = 0.13, mid-p exact binomial method
Statistical Analysis 10: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.06, mid-p exact binomial method
Statistical Analysis 11: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; p = 0.15, mid-p exact binomial method
Statistical Analysis 12: Comparison: 13vPnC; Bronchiolitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.14, mid-p exact binomial method
Statistical Analysis 13: Comparison: 13vPnC; Bronchitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.14, mid-p exact binomial method
Statistical Analysis 14: Comparison: 13vPnC; Bronchospasm: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.14, mid-p exact binomial method
Statistical Analysis 15: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; p = 0.28, mid-p exact binomial method
Statistical Analysis 16: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 14]; Test type: Superiority or Other; p = 0.12, mid-p exact binomial method
Statistical Analysis 17: Comparison: 13vPnC; Constipation: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.68, mid-p exact binomial method
Statistical Analysis 18: Comparison: 13vPnC; Croup: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.24, mid-p exact binomial method
Statistical Analysis 19: Comparison: 13vPnC; Dehydration: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.61, mid-p exact binomial method
Statistical Analysis 20: Comparison: 13vPnC; Dermatitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.28, mid-p exact binomial method
Statistical Analysis 21: Comparison: 13vPnC; Dyspnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.62, mid-p exact binomial method
Statistical Analysis 22: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 20]; Test type: Superiority or Other; p = 0.63, mid-p exact binomial method
Statistical Analysis 23: Comparison: 13vPnC; Fever: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.66, mid-p exact binomial method
Statistical Analysis 24: Comparison: 13vPnC; Fussy infant: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.68, mid-p exact binomial method
Statistical Analysis 25: Comparison: 13vPnC; Gastroenteritis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.18, mid-p exact binomial method
Statistical Analysis 26: Comparison: 13vPnC; [analysis description as in outcome 5, analysis 23]; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 27: Comparison: 13vPnC; Hematoma: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.99, mid-p exact binomial method
Statistical Analysis 28: Comparison: 13vPnC; Hypopotassemia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.25, mid-p exact binomial method
Statistical Analysis 29: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 25]; Test type: Superiority or Other; p = 0.37, mid-p exact binomial method
Statistical Analysis 30: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 26]; Test type: Superiority or Other; p = 0.12, mid-p exact binomial method
Statistical Analysis 31: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 27]; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 32: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 29]; Test type: Superiority or Other; p = 0.25, mid-p exact binomial method
Statistical Analysis 33: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 30]; Test type: Superiority or Other; p = 0.82, mid-p exact binomial method
Statistical Analysis 34: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 31]; Test type: Superiority or Other; p = 0.38, mid-p exact binomial method
Statistical Analysis 35: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 32]; Test type: Superiority or Other; p = 0.78, mid-p exact binomial method
Statistical Analysis 36: Comparison: 13vPnC; Pneumonia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.65, mid-p exact binomial method
Statistical Analysis 37: Comparison: 13vPnC; Rash: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.17, mid-p exact binomial method
Statistical Analysis 38: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 36]; Test type: Superiority or Other; p = 0.22, mid-p exact binomial method
Statistical Analysis 39: Comparison: 13vPnC; Single seizure: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.81, mid-p exact binomial method
Statistical Analysis 40: Comparison: 13vPnC; Stomatitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 41: Comparison: 13vPnC; Stridor: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.13, mid-p exact binomial method
Statistical Analysis 42: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 37]; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 43: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 40]; Test type: Superiority or Other; p = 0.99, mid-p exact binomial method
Statistical Analysis 44: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 41]; Test type: Superiority or Other; p = 0.99, mid-p exact binomial method
Statistical Analysis 45: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 42]; Test type: Superiority or Other; p = 0.25, mid-p exact binomial method
Statistical Analysis 46: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 43]; Test type: Superiority or Other; p = 0.96, mid-p exact binomial method
Statistical Analysis 47: Comparison: 13vPnC; Urticaria: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.97, mid-p exact binomial method
Statistical Analysis 48: Comparison: 13vPnC; Viral syndrome: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.19, mid-p exact binomial method
Statistical Analysis 49: Comparison: 13vPnC; Weakness: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.25, mid-p exact binomial method
Statistical Analysis 50: Comparison: 13vPnC; Wheezing: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.03, mid-p exact binomial method

13. Primary Outcome: Relative Risk of Medically Attended Events Between 30-day Risk Window and 30-day Self-control Window: Primary Series Inpatient
Description: Relative risk for given event = incidence rate (risk window) / incidence rate (self-control window). For primary series (Dose 1, 2, 3 combined), all 30-day risk windows and all post-dose 30-day control windows were summed. Relative risk in inpatient health care setting for primary series was assessed by comparing the combined incidence rate of reported events in inpatient setting per 1000 person-months occurring within 30 days after Dose 1, 2, and 3 (risk window) with the combined self-control period occurring during the subsequent 30 days for each dose (self-control windows after risk window for each dose). Relative risk and exact 2-sided 90% CIs were reported. Medically attended events were documented retrospectively according to ICD-9 coding. Results were reported for events reported in either of the windows.
Time Frame: 30 days after Dose 1, 2, 3 combined (risk window for primary series), 30 days after risk window for Dose 1, 2, 3 combined (post-dose self-control window for primary series)
Population: as for outcome 10
Measure: Number (90% Confidence Interval); unit: ratio
Arm/Group | 13vPnC
Number analyzed (Participants) | 44178
ratio
  Abnormal involuntary movements | 4.69 [1.40 to 21.45]
  Acute bronchiolitis due to RSV | 1.57 [1.12 to 2.23]
  Acute febrile mucocutaneous lymph node syndrome | 3.29 [0.91 to 15.67]
  Acute otitis media | 0.88 [0.47 to 1.63]
  Acute pyelonephritis without RMN lesion | 1.88 [0.76 to 4.94]
  Alkalosis | 6.57 [1.30 to 74.09]
  Apnea | 1.56 [0.67 to 3.84]
  Apparent life threatening event infant | 1.76 [0.86 to 3.75]
  Asthma with acute exacerbation | 2.82 [0.42 to 36.59]
  Asthma, unspecified, unspecified status | 0.80 [0.41 to 1.55]
  Bronchiolitis | 1.55 [1.01 to 2.42]
  Bronchitis | 0.94 [0.15 to 6.00]
  Bronchospasm | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Candidiasis of mouth | 4.22 [1.23 to 19.53]
  Cellulitis and abscess of trunk | 0.94 [0.27 to 3.23]
  Constipation | 0.75 [0.33 to 1.66]
  Croup | 1.13 [0.55 to 2.33]
  Dehydration | 1.17 [0.83 to 1.65]
  Dermatitis | 1.06 [0.47 to 2.41]
  Dyspnea | 0.88 [0.47 to 1.63]
  Failure to thrive | 1.35 [0.86 to 2.12]
  Fever | 1.30 [0.78 to 2.19]
  Fussy infant | 0.94 [0.27 to 3.23]
  Gastroenteritis | 1.17 [0.37 to 3.83]
  Hand, foot and mouth disease | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Hypopotassemia | NA [1.61 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Lipoma of other specified sites | 0.75 [0.23 to 2.36]
  Methicillin susceptible Staphylococcus aureus | 1.41 [0.59 to 3.51]
  Nausea and vomiting | 0.47 [0.03 to 4.04]
  Neonatal bradycardia | NA [1.21 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Other diseases of nasal cavity and sinuses | 0.56 [0.23 to 1.32]
  Other specified cardiac dysrhythmias | 2.82 [1.11 to 8.00]
  Pilonidal cyst without mention of abscess | 1.96 [1.40 to 2.78]
  Pneumonia | 0.94 [0.55 to 1.61]
  Primary apnea of newborn | NA [2.01 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Rash | 0.54 [0.18 to 1.52]
  Respiratory syncytial virus | 0.47 [0.03 to 4.04]
  Retinopathy of prematurity stage 2 | NA [1.21 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Single seizure | 0.61 [0.35 to 1.06]
  Stridor | 1.41 [0.59 to 3.51]
  Subconjunctival hemorrhage | NA [NA to 8.45] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Umbilical hernia without obstruction/gangrene | 2.66 [1.24 to 6.14]
  Unspecified bacterial pneumonia | 2.82 [0.75 to 13.74]
  Unspecified septicemia | 2.19 [0.71 to 7.80]
  Urinary tract infection | 0.88 [0.48 to 1.60]
  Urticaria | NA [NA to 8.45] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Viral syndrome | 0.87 [0.44 to 1.69]
  Weakness | NA [0.81 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Wheezing | 0.94 [0.22 to 4.02]
Statistical Analysis 1: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.03, mid-p exact binomial method
Statistical Analysis 2: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.03, mid-p exact binomial method
Statistical Analysis 3: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.13, mid-p exact binomial method
Statistical Analysis 4: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p = 0.73, mid-p exact binomial method
Statistical Analysis 5: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.26, mid-p exact binomial method
Statistical Analysis 6: Comparison: 13vPnC; Alkalosis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.05, mid-p exact binomial method
Statistical Analysis 7: Comparison: 13vPnC; Apnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.40, mid-p exact binomial method
Statistical Analysis 8: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; p = 0.20, mid-p exact binomial method
Statistical Analysis 9: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.41, mid-p exact binomial method
Statistical Analysis 10: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; p = 0.59, mid-p exact binomial method
Statistical Analysis 11: Comparison: 13vPnC; Bronchiolitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.10, mid-p exact binomial method
Statistical Analysis 12: Comparison: 13vPnC; Bronchitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.95, mid-p exact binomial method
Statistical Analysis 13: Comparison: 13vPnC; Bronchospasm: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 14: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; p = 0.05, mid-p exact binomial method
Statistical Analysis 15: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 14]; Test type: Superiority or Other; p = 0.93, mid-p exact binomial method
Statistical Analysis 16: Comparison: 13vPnC; Constipation: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.56, mid-p exact binomial method
Statistical Analysis 17: Comparison: 13vPnC; Croup: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.79, mid-p exact binomial method
Statistical Analysis 18: Comparison: 13vPnC; Dehydration: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.46, mid-p exact binomial method
Statistical Analysis 19: Comparison: 13vPnC; Dermatitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.92, mid-p exact binomial method
Statistical Analysis 20: Comparison: 13vPnC; Dyspnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.73, mid-p exact binomial method
Statistical Analysis 21: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 20]; Test type: Superiority or Other; p = 0.27, mid-p exact binomial method
Statistical Analysis 22: Comparison: 13vPnC; Fever: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.40, mid-p exact binomial method
Statistical Analysis 23: Comparison: 13vPnC; Fussy infant: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.93, mid-p exact binomial method
Statistical Analysis 24: Comparison: 13vPnC; Gastroenteritis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.82, mid-p exact binomial method
Statistical Analysis 25: Comparison: 13vPnC; [analysis description as in outcome 5, analysis 23]; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 26: Comparison: 13vPnC; Hypopotassemia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.04, mid-p exact binomial method
Statistical Analysis 27: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 25]; Test type: Superiority or Other; p = 0.69, mid-p exact binomial method
Statistical Analysis 28: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 26]; Test type: Superiority or Other; p = 0.53, mid-p exact binomial method
Statistical Analysis 29: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 27]; Test type: Superiority or Other; p = 0.59, mid-p exact binomial method
Statistical Analysis 30: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 28]; Test type: Superiority or Other; p = 0.07, mid-p exact binomial method
Statistical Analysis 31: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 30]; Test type: Superiority or Other; p = 0.27, mid-p exact binomial method
Statistical Analysis 32: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 31]; Test type: Superiority or Other; p = 0.06, mid-p exact binomial method
Statistical Analysis 33: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 32]; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 34: Comparison: 13vPnC; Pneumonia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.85, mid-p exact binomial method
Statistical Analysis 35: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 34]; Test type: Superiority or Other; p = 0.02, mid-p exact binomial method
Statistical Analysis 36: Comparison: 13vPnC; Rash: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.33, mid-p exact binomial method]
Statistical Analysis 37: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 36]; Test type: Superiority or Other; p = 0.59, mid-p exact binomial method
Statistical Analysis 38: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 37]; Test type: Superiority or Other; p = 0.07, mid-p exact binomial method
Statistical Analysis 39: Comparison: 13vPnC; Single seizure: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.14, mid-p exact binomial method
Statistical Analysis 40: Comparison: 13vPnC; Stridor: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.53, mid-p exact binomial method
Statistical Analysis 41: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 37]; Test type: Superiority or Other; p = 0.48, mid-p exact binomial method
Statistical Analysis 42: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 40]; Test type: Superiority or Other; p = 0.03, mid-p exact binomial method
Statistical Analysis 43: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 41]; Test type: Superiority or Other; p = 0.21, mid-p exact binomial method
Statistical Analysis 44: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 42]; Test type: Superiority or Other; p = 0.27, mid-p exact binomial method
Statistical Analysis 45: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 43]; Test type: Superiority or Other; p = 0.73, mid-p exact binomial method
Statistical Analysis 46: Comparison: 13vPnC; Urticaria: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.48, mid-p exact binomial method
Statistical Analysis 47: Comparison: 13vPnC; Viral syndrome: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.73, mid-p exact binomial method
Statistical Analysis 48: Comparison: 13vPnC; Weakness: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.14, mid-p exact binomial method
Statistical Analysis 49: Comparison: 13vPnC; Wheezing: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.94, mid-p exact binomial method

14. Primary Outcome: Relative Risk of Medically Attended Events Between 30-day Risk Window and 30-day Self-control Window: Primary Series Emergency Department
Description: Relative risk for given event = incidence rate (risk window) / incidence rate (self-control window). For primary series (Dose 1, 2, 3 combined), all 30-day risk windows and all post-dose 30-day control windows were summed. Relative risk in emergency department health care setting for primary series was assessed by comparing the combined incidence rate of reported events in emergency department setting per 1000 person-months occurring within 30 days after Dose 1, 2, and 3 (risk window) with the combined self-control period occurring during the subsequent 30 days for each dose (self-control windows after risk window for each dose). Relative risk and exact 2-sided 90% CIs were reported. Medically attended events were documented retrospectively according to ICD-9 coding. Results were reported for events reported in either of the windows.
Time Frame: as for outcome 13
Population: as for outcome 10
Measure: Number (90% Confidence Interval); unit: ratio
Arm/Group | 13vPnC
Number analyzed (Participants) | 44178
ratio
  Abnormal involuntary movements | 1.56 [0.46 to 5.92]
  Acute bronchiolitis due to RSV | 1.27 [0.78 to 2.08]
  Acute febrile mucocutaneous lymph node syndrome | NA [NA to 8.45] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Acute otitis media | 0.73 [0.59 to 0.89]
  Acute pyelonephritis without RMN lesion | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Adverse drug reaction | 0.94 [0.27 to 3.23]
  Alkalosis | NA [0.10 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Apnea | 1.88 [0.68 to 5.62]
  Apparent life threatening event infant | 1.74 [0.81 to 3.93]
  Asthma with acute exacerbation | 2.82 [0.42 to 36.59]
  Asthma, unspecified, unspecified status | 0.63 [0.41 to 0.95]
  Bronchiolitis | 0.89 [0.74 to 1.07]
  Bronchitis | 0.70 [0.33 to 1.47]
  Bronchospasm | 1.20 [0.77 to 1.88]
  Candidiasis of mouth | 0.67 [0.24 to 1.79]
  Cellulitis and abscess of trunk | NA [NA to 8.45] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Constipation | 0.81 [0.52 to 1.27]
  Croup | 0.95 [0.75 to 1.19]
  Dehydration | 0.96 [0.66 to 1.40]
  Dermatitis | 0.56 [0.34 to 0.92]
  Dyspnea | 1.37 [0.89 to 2.13]
  Failure to thrive | 3.76 [0.63 to 45.97]
  Fever | 1.17 [1.04 to 1.31]
  Fussy infant | 1.17 [0.87 to 1.58]
  Gastroenteritis | 0.73 [0.50 to 1.06]
  Hand, foot and mouth disease | 1.13 [0.40 to 3.23]
  Hematoma | 0.70 [0.18 to 2.62]
  Nausea and vomiting | 0.86 [0.71 to 1.03]
  Neonatal candida infection | 5.63 [1.07 to 64.71]
  Other diseases of nasal cavity and sinuses | 1.10 [0.79 to 1.54]
  Other specified cardiac dysrhythmias | 1.88 [0.22 to 27.21]
  Pneumonia | 0.85 [0.66 to 1.10]
  Rash | 0.78 [0.56 to 1.09]
  Respiratory syncytial virus | 1.02 [0.51 to 2.07]
  Single seizure | 1.15 [0.68 to 1.95]
  Stomatitis | NA [NA to 2.03] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Stridor | 4.69 [0.85 to 55.34]
  Subconjunctival hemorrhage | NA [1.21 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Umbilical hernia without obstruction/gangrene | 1.41 [0.29 to 7.94]
  Unspecified septicemia | 0.75 [0.23 to 2.36]
  Urinary tract infection | 1.62 [1.17 to 2.26]
  Urticaria | 0.90 [0.54 to 1.49]
  Vaccines adverse reaction | NA [1.21 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Viral syndrome | 0.66 [0.52 to 0.82]
  Weakness | NA [1.21 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window.
  Wheezing | 1.08 [0.76 to 1.53]
Statistical Analysis 1: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.56, mid-p exact binomial method
Statistical Analysis 2: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.43, mid-p exact binomial method
Statistical Analysis 3: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.48, mid-p exact binomial method
Statistical Analysis 4: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p = 0.01, mid-p exact binomial method
Statistical Analysis 5: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 6: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.93, mid-p exact binomial method
Statistical Analysis 7: Comparison: 13vPnC; Alkalosis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 8: Comparison: 13vPnC; Apnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.32, mid-p exact binomial method
Statistical Analysis 9: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; p = 0.24, mid-p exact binomial method
Statistical Analysis 10: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.41, mid-p exact binomial method
Statistical Analysis 11: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; p = 0.06, mid-p exact binomial method
Statistical Analysis 12: Comparison: 13vPnC; Bronchiolitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.31, mid-p exact binomial method
Statistical Analysis 13: Comparison: 13vPnC; Bronchitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.43, mid-p exact binomial method
Statistical Analysis 14: Comparison: 13vPnC; Bronchospasm: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.50, mid-p exact binomial method
Statistical Analysis 15: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; p = 0.51, mid-p exact binomial method
Statistical Analysis 16: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 14]; Test type: Superiority or Other; p = 0.48, mid-p exact binomial method
Statistical Analysis 17: Comparison: 13vPnC; Constipation: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.44, mid-p exact binomial method
Statistical Analysis 18: Comparison: 13vPnC; Croup: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.70, mid-p exact binomial method
Statistical Analysis 19: Comparison: 13vPnC; Dehydration: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.87, mid-p exact binomial method
Statistical Analysis 20: Comparison: 13vPnC; Dermatitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.05, mid-p exact binomial method
Statistical Analysis 21: Comparison: 13vPnC; Dyspnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.24, mid-p exact binomial method
Statistical Analysis 22: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 20]; Test type: Superiority or Other; p = 0.24, mid-p exact binomial method
Statistical Analysis 23: Comparison: 13vPnC; Fever: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.03, mid-p exact binomial method
Statistical Analysis 24: Comparison: 13vPnC; Fussy infant: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.37, mid-p exact binomial method
Statistical Analysis 25: Comparison: 13vPnC; Gastroenteritis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.16, mid-p exact binomial method
Statistical Analysis 26: Comparison: 13vPnC; [analysis description as in outcome 5, analysis 23]; Test type: Superiority or Other; p = 0.85, mid-p exact binomial method
Statistical Analysis 27: Comparison: 13vPnC; Hematoma: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.67, mid-p exact binomial method
Statistical Analysis 28: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 27]; Test type: Superiority or Other; p = 0.18, mid-p exact binomial method
Statistical Analysis 29: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 29]; Test type: Superiority or Other; p = 0.08, mid-p exact binomial method
Statistical Analysis 30: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 30]; Test type: Superiority or Other; p = 0.63, mid-p exact binomial method
Statistical Analysis 31: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 31]; Test type: Superiority or Other; p = 0.66, mid-p exact binomial method
Statistical Analysis 32: Comparison: 13vPnC; Pneumonia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.31, mid-p exact binomial method
Statistical Analysis 33: Comparison: 13vPnC; Rash: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.22, mid-p exact binomial method
Statistical Analysis 34: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 36]; Test type: Superiority or Other; p = 0.96, mid-p exact binomial method
Statistical Analysis 35: Comparison: 13vPnC; Single seizure: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.67, mid-p exact binomial method
Statistical Analysis 36: Comparison: 13vPnC; Stomatitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.23, mid-p exact binomial method
Statistical Analysis 37: Comparison: 13vPnC; Stridor: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.14, mid-p exact binomial method
Statistical Analysis 38: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 37]; Test type: Superiority or Other; p = 0.07, mid-p exact binomial method
Statistical Analysis 39: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 40]; Test type: Superiority or Other; p = 0.74, mid-p exact binomial method
Statistical Analysis 40: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 42]; Test type: Superiority or Other; p = 0.69, mid-p exact binomial method
Statistical Analysis 41: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 43]; Test type: Superiority or Other; p = 0.01, mid-p exact binomial method
Statistical Analysis 42: Comparison: 13vPnC; Urticaria: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.72, mid-p exact binomial method
Statistical Analysis 43: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 42]; Test type: Superiority or Other; p = 0.07, mid-p exact binomial method
Statistical Analysis 44: Comparison: 13vPnC; Viral syndrome: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 45: Comparison: 13vPnC; Weakness: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.07, mid-p exact binomial method
Statistical Analysis 46: Comparison: 13vPnC; Wheezing: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.73, mid-p exact binomial method

15. Primary Outcome: Relative Risk of Medically Attended Events Between 30-day Risk Window and 30-day Self-control Window: Primary Series Inpatient and Emergency Department Combined
Description: Relative risk for given event = incidence rate (risk window) / incidence rate (self-control window). For primary series (Dose 1, 2, 3 combined), all 30-day risk windows and all post-dose 30-day control windows were summed. Relative risk in in inpatient and emergency department health care setting for primary series was assessed by comparing the combined incidence rate of reported events in both the settings per 1000 person-months occurring within 30 days after Dose 1, 2, and 3 (risk window) with the combined self-control period occurring during the subsequent 30 days for each dose (self-control windows after risk window for each dose). Relative risk and exact 2-sided 90% CIs were reported. Medically attended events were documented retrospectively according to ICD-9 coding. Results were reported for events reported in either of the windows.
Time Frame: as for outcome 13
Population: as for outcome 10
Measure: Number (90% Confidence Interval); unit: ratio
Arm/Group | 13vPnC
Number analyzed (Participants) | 44178
ratio
  Abnormal involuntary movements | 2.82 [1.23 to 7.07]
  Acute bronchiolitis due to RSV | 1.50 [1.12 to 2.01]
  Acute febrile mucocutaneous lymph node syndrome | 2.19 [0.71 to 7.80]
  Acute otitis media | 0.75 [0.62 to 0.92]
  Acute pyelonephritis without RMN lesion | 2.07 [0.86 to 5.36]
  Adverse drug reaction | 0.94 [0.27 to 3.23]
  Alkalosis | 6.57 [1.30 to 74.09]
  Apnea | 1.31 [0.66 to 2.66]
  Apparent life threatening event infant | 1.64 [0.91 to 3.04]
  Asthma with acute exacerbation | 2.82 [0.75 to 13.74]
  Asthma, unspecified, unspecified status | 0.65 [0.45 to 0.93]
  Bronchiolitis | 0.95 [0.80 to 1.13]
  Bronchitis | 0.74 [0.37 to 1.44]
  Bronchospasm | 1.24 [0.80 to 1.93]
  Candidiasis of mouth | 1.36 [0.66 to 2.84]
  Cellulitis and abscess of trunk | 0.75 [0.23 to 2.36]
  Constipation | 0.77 [0.52 to 1.14]
  Croup | 0.95 [0.76 to 1.19]
  Dehydration | 0.99 [0.76 to 1.30]
  Dermatitis | 0.68 [0.44 to 1.04]
  Dyspnea | 1.13 [0.79 to 1.62]
  Failure to thrive | 1.43 [0.92 to 2.24]
  Fever | 1.16 [1.03 to 1.29]
  Fussy infant | 1.14 [0.86 to 1.52]
  Gastroenteritis | 0.77 [0.54 to 1.09]
  Hand, foot and mouth disease | 1.31 [0.49 to 3.66]
  Hematoma | 0.70 [0.18 to 2.62]
  Hypopotassemia | NA [1.61 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window
  Lipoma of other specified sites | 0.75 [0.23 to 2.36]
  Methicillin susceptible Staphylococcus aureus | 1.41 [0.59 to 3.51]
  Nausea and vomiting | 0.85 [0.71 to 1.03]
  Neonatal bradycardia | NA [1.21 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window
  Neonatal candida infection | 5.63 [1.07 to 64.71]
  Other diseases of nasal cavity and sinuses | 1.01 [0.74 to 1.37]
  Other specified cardiac dysrhythmias | 3.05 [1.22 to 8.59]
  Pilonidal cyst without mention of abscess | 1.96 [1.40 to 2.78]
  Pneumonia | 0.83 [0.66 to 1.06]
  Primary apnea of newborn | NA [2.01 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window
  Rash | 0.76 [0.55 to 1.05]
  Respiratory syncytial virus | 0.94 [0.49 to 1.81]
  Retinopathy of prematurity stage 2 | NA [1.21 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window
  Single seizure | 0.86 [0.58 to 1.28]
  Stomatitis | NA [NA to 2.03] — Relative risk and lower CI was not estimated because no event was reported during the 30-day risk window.
  Stridor | 1.74 [0.81 to 3.93]
  Subconjunctival hemorrhage | 3.76 [0.63 to 45.97]
  Umbilical hernia without obstruction/gangrene | 2.35 [1.19 to 4.85]
  Unspecified bacterial pneumonia | 2.82 [0.75 to 13.74]
  Unspecified septicemia | 1.72 [0.75 to 4.17]
  Urinary tract infection | 1.39 [1.04 to 1.86]
  Urticaria | 0.86 [0.52 to 1.41]
  Vaccines adverse reaction | NA [1.21 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window
  Viral syndrome | 0.67 [0.54 to 0.83]
  Weakness | NA [1.61 to NA] — Relative risk and upper CI was not estimated because no event was reported during the 30-day self-control window
  Wheezing | 1.09 [0.77 to 1.54]
Statistical Analysis 1: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.04, mid-p exact binomial method
Statistical Analysis 2: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.02, mid-p exact binomial method
Statistical Analysis 3: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.27, mid-p exact binomial method
Statistical Analysis 4: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p = 0.02, mid-p exact binomial method
Statistical Analysis 5: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.18, mid-p exact binomial method
Statistical Analysis 6: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.93, mid-p exact binomial method
Statistical Analysis 7: Comparison: 13vPnC; Alkalosis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.05, mid-p exact binomial method
Statistical Analysis 8: Comparison: 13vPnC; Apnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.52, mid-p exact binomial method
Statistical Analysis 9: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; p = 0.17, mid-p exact binomial method
Statistical Analysis 10: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.21, mid-p exact binomial method
Statistical Analysis 11: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; p = 0.05, mid-p exact binomial method
Statistical Analysis 12: Comparison: 13vPnC; Bronchiolitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.63, mid-p exact binomial method
Statistical Analysis 13: Comparison: 13vPnC; Bronchitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.46, mid-p exact binomial method
Statistical Analysis 14: Comparison: 13vPnC; Bronchospasm: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.42, mid-p exact binomial method
Statistical Analysis 15: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; p = 0.49, mid-p exact binomial method
Statistical Analysis 16: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 14]; Test type: Superiority or Other; p = 0.69, mid-p exact binomial method
Statistical Analysis 17: Comparison: 13vPnC; Constipation: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.28, mid-p exact binomial method
Statistical Analysis 18: Comparison: 13vPnC; Croup: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.69, mid-p exact binomial method
Statistical Analysis 19: Comparison: 13vPnC; Dehydration: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.95, mid-p exact binomial method
Statistical Analysis 20: Comparison: 13vPnC; Dermatitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.13, mid-p exact binomial method
Statistical Analysis 21: Comparison: 13vPnC; Dyspnea: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.57, mid-p exact binomial method
Statistical Analysis 22: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 20]; Test type: Superiority or Other; p = 0.18, mid-p exact binomial method
Statistical Analysis 23: Comparison: 13vPnC; Fever: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.03, mid-p exact binomial method
Statistical Analysis 24: Comparison: 13vPnC; Fussy infant: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.45, mid-p exact binomial method
Statistical Analysis 25: Comparison: 13vPnC; Gastroenteritis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.21, mid-p exact binomial method
Statistical Analysis 26: Comparison: 13vPnC; [analysis description as in outcome 5, analysis 23]; Test type: Superiority or Other; p = 0.66, mid-p exact binomial method
Statistical Analysis 27: Comparison: 13vPnC; Hematoma: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.67, mid-p exact binomial method
Statistical Analysis 28: Comparison: 13vPnC; Hypopotassemia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.04, mid-p exact binomial method
Statistical Analysis 29: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 25]; Test type: Superiority or Other; p = 0.69, mid-p exact binomial method
Statistical Analysis 30: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 26]; Test type: Superiority or Other; p = 0.53, mid-p exact binomial method
Statistical Analysis 31: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 27]; Test type: Superiority or Other; p = 0.16, mid-p exact binomial method
Statistical Analysis 32: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 28]; Test type: Superiority or Other; p = 0.07, mid-p exact binomial method
Statistical Analysis 33: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 29]; Test type: Superiority or Other; p = 0.08, mid-p exact binomial method
Statistical Analysis 34: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 30]; Test type: Superiority or Other; p = 0.98, mid-p exact binomial method
Statistical Analysis 35: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 31]; Test type: Superiority or Other; p = 0.04, mid-p exact binomial method
Statistical Analysis 36: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 32]; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 37: Comparison: 13vPnC; Pneumonia: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.22, mid-p exact binomial method
Statistical Analysis 38: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 34]; Test type: Superiority or Other; p = 0.02, mid-p exact binomial method
Statistical Analysis 39: Comparison: 13vPnC; Rash: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.17, mid-p exact binomial method
Statistical Analysis 40: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 36]; Test type: Superiority or Other; p = 0.87, mid-p exact binomial method
Statistical Analysis 41: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 37]; Test type: Superiority or Other; p = 0.07, mid-p exact binomial method
Statistical Analysis 42: Comparison: 13vPnC; Single seizure: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.54, mid-p exact binomial method
Statistical Analysis 43: Comparison: 13vPnC; Stomatitis: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.23, mid-p exact binomial method
Statistical Analysis 44: Comparison: 13vPnC; Stridor: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.24, mid-p exact binomial method
Statistical Analysis 45: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 37]; Test type: Superiority or Other; p = 0.24, mid-p exact binomial method
Statistical Analysis 46: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 40]; Test type: Superiority or Other; p = 0.04, mid-p exact binomial method
Statistical Analysis 47: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 41]; Test type: Superiority or Other; p = 0.21, mid-p exact binomial method
Statistical Analysis 48: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 42]; Test type: Superiority or Other; p = 0.29, mid-p exact binomial method
Statistical Analysis 49: Comparison: 13vPnC; [analysis description as in outcome 1, analysis 43]; Test type: Superiority or Other; p = 0.06, mid-p exact binomial method
Statistical Analysis 50: Comparison: 13vPnC; Urticaria: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.61, mid-p exact binomial method
Statistical Analysis 51: Comparison: 13vPnC; [analysis description as in outcome 2, analysis 42]; Test type: Superiority or Other; p = 0.07, mid-p exact binomial method
Statistical Analysis 52: Comparison: 13vPnC; Viral syndrome: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p < 0.01, mid-p exact binomial method
Statistical Analysis 53: Comparison: 13vPnC; Weakness: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.04, mid-p exact binomial method
Statistical Analysis 54: Comparison: 13vPnC; Wheezing: p-value was estimated using the mid-p exact binomial method. The null hypothesis was relative risk = 1; Test type: Superiority or Other; p = 0.68, mid-p exact binomial method

ADVERSE EVENTS:
Description: Adverse events (AEs) and serious adverse events (SAEs) were not planned to be collected as this was a non-interventional, observational study, consisting of secondary analysis of de-identified electronic health care database and coded data which did not meet the criteria for reportable AEs.
Arm/Group | 13vPnC
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.